CLINICAL TRIAL: NCT04852978
Title: A Phase 2 Randomized, Open-Label, Parallel Group Study to Assess the Immunogenicity, Safety, and Tolerability of Moderna mRNA-1273 Vaccine Administered With Casirivimab+Imdevimab in Healthy Adult Volunteers
Brief Title: COVID-19 Study to Assess Immunogenicity, Safety, and Tolerability of Moderna mRNA-1273 Vaccine Administered With Casirivimab+Imdevimab in Healthy Adult Volunteers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R10933-10987-COV-2118
Record Dates: First submitted 2021-04-19; First posted 2021-04-21 (Actual); Results first posted 2024-08-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Healthy; Chronic Stable Illness
MeSH Terms: interventions — casirivimab and imdevimab drug combination; casirivimab; imdevimab; 2019-nCoV Vaccine mRNA-1273

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- Wave 1 Dose 1 (Experimental)
  Interventions: Drug: casirivimab+imdevimab; Biological: Moderna mRNA-1273 vaccine
- Wave 1 Dose 2 (Experimental)
  Interventions: Drug: casirivimab+imdevimab; Biological: Moderna mRNA-1273 vaccine
- Wave 1 Dose 3 (Experimental)
  Interventions: Drug: casirivimab+imdevimab; Biological: Moderna mRNA-1273 vaccine
- Wave 1 Vaccine only (Experimental)
  Interventions: Biological: Moderna mRNA-1273 vaccine
- Wave 2 Dose 1 (Experimental)
  Interventions: Drug: casirivimab+imdevimab; Biological: Moderna mRNA-1273 vaccine
- Wave 2 Dose 2 (Experimental)
  Interventions: Drug: casirivimab+imdevimab; Biological: Moderna mRNA-1273 vaccine
- Wave 2 Vaccine only (Experimental)
  Interventions: Biological: Moderna mRNA-1273 vaccine
- Wave 3 Dose 1 (Experimental)
  Interventions: Drug: casirivimab+imdevimab; Biological: Moderna mRNA-1273 vaccine
- Wave 3 Dose 2 (Experimental)
  Interventions: Drug: casirivimab+imdevimab; Biological: Moderna mRNA-1273 vaccine
- Wave 3 Vaccine only (Experimental)
  Interventions: Biological: Moderna mRNA-1273 vaccine
- Wave 4 Dose 1 (Experimental)
  Interventions: Drug: casirivimab+imdevimab; Biological: Moderna mRNA-1273 vaccine
- Wave 4 Vaccine only (Experimental)
  Interventions: Biological: Moderna mRNA-1273 vaccine

INTERVENTIONS:
Drug: casirivimab+imdevimab — Wave 1 Intravenous (IV) administration Wave 2 Subcutaneous administration
  Other Names: REGN10933; REGN10987; REGN-COV2; REGEN-COV™; Ronapreve™
  Arms: Wave 1 Dose 1; Wave 1 Dose 2; Wave 1 Dose 3; Wave 2 Dose 1; Wave 2 Dose 2; Wave 3 Dose 1; Wave 3 Dose 2; Wave 4 Dose 1
Biological: Moderna mRNA-1273 vaccine — Single intramuscular (IM) injection

SUMMARY:
The primary objectives of the study are:

* To evaluate the extent of effect, if any, of REGN10933+REGN10987 administration on vaccine-induced neutralizing antibody responses to SARS-CoV-2 by Moderna mRNA-1273
* To evaluate the time interval required between REGN10933+REGN10987 administration and Moderna mRNA-1273 vaccination, to ensure no meaningful impact on vaccine-induced neutralizing antibody responses to SARS-CoV-2

The secondary objectives of the study are:

* To quantify the alteration of antigen specificity of vaccine-induced SARS-CoV-2 antibody responses when administered with different dose regimens of REGN10933+REGN10987
* To evaluate the safety and tolerability of REGN10933+REGN10987 and Moderna mRNA-1273 vaccine when administered in close succession
* To assess the concentrations of REGN10933 and REGN10987 in serum over time in participants who receive REGN10933+REGN10987 and Moderna mRNA-1273 vaccine
* To evaluate the immunogenicity of REGN10933 and REGN10987 over time

ELIGIBILITY:
Key Inclusion Criteria:

1. Healthy or has chronic medical condition(s) that are stable and well-controlled in the opinion of the investigator and that are not likely to require significant medical intervention through the end of study
2. Willing and able to comply with study visits and study-related procedures, including compliance with site precautionary requirements related to SARS-CoV-2 infection and transmission

Key Exclusion Criteria:

1. Positive RT-PCR test result for SARS-CoV-2 infection at screening or baseline
2. Positive serology test result for anti-SARS-CoV-2 antibodies at screening or baseline
3. COVID-19 diagnosis, positive SARS-CoV-2 infection, or positive SARS-CoV-2 serology at any time prior to screening
4. Previously received an investigational, authorized, or approved coronavirus vaccine (eg, SARS-CoV-2 vaccine, MERS-CoV vaccine)
5. Currently enrolled in, or has plans to enroll in, any interventional study to prevent or treat COVID-19
6. Received investigational or approved passive antibodies for SARS-CoV-2 infection prophylaxis ad defined in the protocol
7. Received intravenous immunoglobulin (IVIG) or blood products in the last 3 months
8. Any physical examination findings and/or history of any illness that, in the opinion of the study investigator, might confound the results of the study or pose an additional risk to the subject by study participation
9. History of clinically significant cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, psychiatric or neurological disease, as assessed by the investigator, that may confound the results of the study or pose an additional risk to the subject by study participation
10. Medically attended acute illness or hospitalization (ie, >24 hours) for any reason within 30 days prior to screening
11. Clinical history of myocarditis and/or pericarditis

Note: Other protocol-defined Inclusion/ Exclusion Criteria apply

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 295 (Actual)
Dates: Start 2021-04-29 (Actual); Primary Completion 2022-11-21 (Actual); Study Completion 2022-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (6):
- United States (6):
  - Regeneron Research Site, Little Rock, Arkansas
  - Regeneron Research Site, Rogers, Arkansas
  - Regeneron Research Site, Hialeah, Florida
  - Regeneron Research Site, Miami, Florida
  - Regeneron Research Site, Orlando, Florida
  - Regeneron Research Site, Dayton, Ohio

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication, has made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry), has the legal authority to share the data, and has ensured the ability to protect participant privacy.
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/

REFERENCES:
- [Derived] Isa F, Gonzalez Ortiz AM, Meyer J, Hamilton JD, Olenchock BA, Brackin T, Ganguly S, Forleo-Neto E, Faria L, Heirman I, Marovich M, Hutter J, Polakowski L, Irvin SC, Thakur M, Hooper AT, Baum A, Petro CD, Fakih FA, McElrath MJ, De Rosa SC, Cohen KW, Williams LD, Hellman CA, Odeh AJ, Patel AH, Tomaras GD, Geba GP, Kyratsous CA, Musser B, Yancopoulos GD, Herman GA; Trial Working Group. Effect of timing of casirivimab and imdevimab administration relative to mRNA-1273 COVID-19 vaccination on vaccine-induced SARS-CoV-2 neutralising antibody responses: a prospective, open-label, phase 2, randomised controlled trial. Lancet Infect Dis. 2025 Jan;25(1):52-67. doi: 10.1016/S1473-3099(24)00421-3. Epub 2024 Sep 2. PMID 39236733

RESULTS

PARTICIPANT FLOW:
Groups:
- Vaccine Only: Vaccine only, no study drug
- REGN10933+REGN10987 + Vaccine 1200 mg Day 1 IV: REGN10933+REGN10987 + Vaccine 1200 mg Day 1 IV
- REGN10933+REGN10987 + Vaccine 300 mg Day 1 IV: REGN10933+REGN10987 + Vaccine 300 mg Day 1 IV
- REGN10933+REGN10987 + Vaccine 150 mg Day 1 IV: REGN10933+REGN10987 + Vaccine 150 mg Day 1 IV
- REGN10933+REGN10987 + Vaccine 48 mg Day 1 IV: REGN10933+REGN10987 + Vaccine 48 mg Day 1 IV
- REGN10933+REGN10987 + Vaccine 12 mg Day 1 IV: REGN10933+REGN10987 + Vaccine 12 mg Day 1 IV
- REGN10933+REGN10987 + Vaccine 1200 mg Day 7 IV: REGN10933+REGN10987 + Vaccine 1200 mg Day 7 IV
- REGN10933+REGN10987 + Vaccine 1200 mg Day 1 SC: REGN10933+REGN10987 + Vaccine 1200 mg Day 1 SC
- REGN10933+REGN10987 + Vaccine 600 mg Day 1 SC: REGN10933+REGN10987 + Vaccine 600 mg Day 1 SC
Period: Overall Study
Arm/Group | Vaccine Only | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 300 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 150 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 48 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 12 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 7 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 SC | REGN10933+REGN10987 + Vaccine 600 mg Day 1 SC
Started | 48 | 28 | 29 | 28 | 33 | 31 | 26 | 35 | 35
Completed | 41 | 23 | 24 | 27 | 26 | 24 | 22 | 29 | 32
Not Completed | 7 | 5 | 5 | 1 | 7 | 7 | 4 | 6 | 3
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Sponsor request | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 3 | 2 | 2 | 0 | 2 | 4 | 1 | 2 | 2
Not completed — Withdrawal by Subject | 4 | 2 | 2 | 1 | 5 | 3 | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Population: The safety analysis set (SAF) includes all randomized subjects who have been vaccinated with at least one dose or received any study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | Vaccine Only | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 300 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 150 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 48 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 12 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 7 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 SC | REGN10933+REGN10987 + Vaccine 600 mg Day 1 SC | Total
Number analyzed (Participants) | 48 | 28 | 29 | 28 | 33 | 31 | 26 | 35 | 35 | 293
Age, Customized [Mean (Standard Deviation); unit: years] | 40.2 (12.17) | 41.8 (13.98) | 39.3 (12.76) | 39.7 (13.50) | 41.6 (12.73) | 41.1 (11.23) | 39.8 (13.76) | 43.8 (12.99) | 46.3 (11.53) | 41.6 (12.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 13 | 9 | 13 | 17 | 16 | 14 | 14 | 19 | 143
  Male | 20 | 15 | 20 | 15 | 16 | 15 | 12 | 21 | 16 | 150
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 9 | 12 | 9 | 16 | 19 | 17 | 11 | 12 | 121
  Not Hispanic or Latino | 31 | 19 | 17 | 19 | 17 | 12 | 9 | 24 | 23 | 171
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 3
  Asian | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Black or African American | 16 | 10 | 7 | 9 | 9 | 7 | 7 | 10 | 7 | 82
  White | 32 | 18 | 22 | 18 | 23 | 21 | 19 | 24 | 27 | 204
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: 50% Inhibitory Dilution (ID50) Titers of Vaccine-induced Neutralizing Antibodies to the SARS-CoV-2 S Protein in Individuals Who Received High Dose REGN10933+REGN10987 (1200 mg)
Description: High dose - (1200 mg arms)
Time Frame: 56 days after first dose of vaccine
Population: Per protocol set (PPS) includes all randomized participants who have received both doses of vaccine and who do not meet the exclusion criteria. The PPS is the primary analysis set for assessing vaccine response related endpoints.
Measure: Mean (Standard Deviation); unit: Titer
Arm/Group | Vaccine Only | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 SC | REGN10933+REGN10987 + Vaccine 1200 mg Day 7 IV
Number analyzed (Participants) | 41 | 24 | 32 | 22
Titer | 2594.9 (1981.5) | 1818.6 (2365.8) | 980.8 (1015.1) | 2576.8 (2736.1)

2. Primary Outcome: 50% Inhibitory Dilution (ID50) Titers of Vaccine-induced Neutralizing Antibodies to the SARS-CoV-2 S Protein in Individual Who Received Submaximal Dose Levels of REGN10933+REGN10987 (Less Than 1200 mg)
Description: Submaximal dose - (150 mg, 300 mg, 600 mg, 48 mg, and 12 mg)
Time Frame: 56 days after first dose of vaccine
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Titer
Arm/Group | Vaccine Only | REGN10933+REGN10987 + Vaccine 300 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 150 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 48 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 12 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 600 mg Day 1 SC
Number analyzed (Participants) | 41 | 26 | 26 | 28 | 24 | 31
Titer | 2594.9 (1981.5) | 780.8 (771.1) | 716.1 (664.9) | 4922.8 (11157.3) | 2422.2 (2882.7) | 1549.5 (4334.1)

3. Secondary Outcome: Absolute Values in Concentrations of Vaccine-induced Antibodies to SARS-CoV-2 Antigens Over Time (S1-RBD IgA)
Description: Anti-S1-RBD protein
Time Frame: Up to 365 Days from 1st dose of Vaccination
Population: Per protocol set (PPS) includes all randomized participants who have received both doses of vaccine and who do not meet the exclusion criteria. The PPS is the primary analysis set for assessing vaccine response related endpoints. As was pre-specified in the study protocol, only participants in the "Vaccine Only" and " REGN10933+REGN10987 + Vaccine 1200 mg Day 7" Arm/Group were assessed for measure 6 days after the first vaccine.
Measure: Mean (Standard Deviation); unit: Binding Antibody Unit (BAU)/mL
Arm/Group | Vaccine Only | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 300 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 150 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 48 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 12 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 7 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 SC | REGN10933+REGN10987 + Vaccine 600 mg Day 1 SC
Number analyzed (Participants) | 42 | 26 | 26 | 26 | 28 | 24 | 24 | 32 | 32
Binding Antibody Unit (BAU)/mL
  Baseline: number analyzed (Participants) | 41 | 26 | 26 | 26 | 28 | 24 | 23 | 32 | 32
  Baseline | 18.7 (9.2) | 15.7 (0.0) | 20.7 (25.2) | 15.7 (0.0) | 20.1 (11.6) | 24.4 (22.5) | 22.6 (14.4) | 20.2 (11.2) | 17.6 (10.5)
  6 Days after 1st Vaccine: number analyzed (Participants) | 5 | 0 | 0 | 00 | 0 | 0 | 24 | 0 | 0
  6 Days after 1st Vaccine | 47.5 (31.8) |  |  |  |  |  | 352.9 (1590.7) |  |
  14 Days after 1st Vaccine: number analyzed (Participants) | 42 | 26 | 25 | 25 | 28 | 24 | 24 | 31 | 32
  14 Days after 1st Vaccine | 1176.5 (1758.5) | 884.0 (860.0) | 1510.6 (2141.5) | 730.4 (963.2) | 638.6 (662.1) | 673.7 (871.0) | 1046.0 (1726.3) | 1184.6 (1716.7) | 902.0 (1485.9)
  28 Days after 1st Vaccine | 373.0 (416.1) | 276.3 (461.4) | 297.8 (514.2) | 171.9 (193.1) | 209.0 (207.0) | 246.0 (451.3) | 592.3 (1587.1) | 351.0 (566.1) | 259.4 (520.4)
  42 Days after 1st Vaccine: number analyzed (Participants) | 41 | 25 | 26 | 26 | 28 | 21 | 20 | 32 | 31
  42 Days after 1st Vaccine | 2610.7 (2032.3) | 2318.5 (2387.2) | 2190.4 (2163.5) | 2022.8 (2170.3) | 1989.5 (1797.0) | 1246.5 (1017.9) | 1460.5 (1724.8) | 1714.4 (1779.3) | 1763.1 (1444.0)
  56 Days after 1st Vaccine: number analyzed (Participants) | 41 | 24 | 26 | 26 | 28 | 22 | 22 | 32 | 31
  56 Days after 1st Vaccine | 1327.7 (1497.7) | 1146.2 (1738.7) | 769.1 (836.1) | 845.9 (1056.3) | 787.9 (630.1) | 669.4 (813.7) | 841.7 (1587.0) | 889.6 (1475.2) | 732.0 (785.6)
  168 Days after 1st Vaccine: number analyzed (Participants) | 40 | 24 | 25 | 26 | 25 | 22 | 21 | 31 | 31
  168 Days after 1st Vaccine | 1825.0 (2690.3) | 986.3 (1718.1) | 358.8 (610.3) | 1211.0 (2194.5) | 1772.6 (2353.2) | 871.1 (1584.9) | 3053.1 (3077.9) | 715.2 (1658.4) | 346.2 (888.1)
  252 Days after 1st Vaccine: number analyzed (Participants) | 37 | 24 | 24 | 26 | 22 | 18 | 20 | 27 | 30
  252 Days after 1st Vaccine | 3665.4 (3141.0) | 3488.8 (3126.5) | 3180.0 (3171.6) | 3174.7 (2840.8) | 1508.8 (1831.0) | 1539.2 (1681.9) | 2898.1 (2674.8) | 4269.9 (3316.2) | 3556.1 (3122.6)
  365 Days after 1st Vaccine: number analyzed (Participants) | 37 | 22 | 23 | 26 | 23 | 18 | 20 | 27 | 30
  365 Days after 1st Vaccine | 2722.7 (2680.0) | 3904.4 (3036.1) | 2804.1 (2533.8) | 3008.7 (2609.0) | 2180.7 (1934.9) | 2155.8 (2369.2) | 2727.5 (2632.9) | 3193.5 (2890.2) | 3136.9 (2864.3)

4. Secondary Outcome: Median Fold Change of Concentrations of Vaccine-induced Antibodies to SARS-CoV-2 Antigens Over Time (S1-RBD IgA)
Description: Anti-S1-RBD protein. Fold Change based on medians = (median value in vaccine only arm / median value in the active arm)
Time Frame: Up to 365 Days from 1st dose of Vaccination
Population: Per protocol set (PPS) includes all randomized participants who have received both doses of vaccine and who do not meet the exclusion criteria. The PPS is the primary analysis set for assessing vaccine response related endpoints. As was pre-specified in the study protocol, only participants in the "Vaccine Only" and " REGN10933+REGN10987 + Vaccine 1200 mg Day 7" Arm/Group were assessed for measure 6 days after the first vaccine,
Measure: Number; unit: Fold Change
Arm/Group | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 300 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 150 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 48 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 12 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 7 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 SC | REGN10933+REGN10987 + Vaccine 600 mg Day 1 SC
Number analyzed (Participants) | 26 | 26 | 26 | 28 | 24 | 24 | 32 | 32
Fold Change
  6 Days after 1st Vaccine: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 24 | 0 | 0
  6 Days after 1st Vaccine |  |  |  |  |  | 3.2 |  |
  14 Days after 1st Vaccine: number analyzed (Participants) | 26 | 25 | 25 | 28 | 24 | 24 | 31 | 32
  14 Days after 1st Vaccine | 0.8 | 0.6 | 1.6 | 1.1 | 1.9 | 1.3 | 1.0 | 1.3
  28 Days after 1st Vaccine | 1.7 | 2.0 | 2.6 | 1.9 | 2.7 | 1.7 | 1.4 | 2.4
  42 Days after 1st Vaccine: number analyzed (Participants) | 25 | 26 | 26 | 28 | 21 | 20 | 32 | 31
  42 Days after 1st Vaccine | 1.5 | 1.6 | 1.7 | 1.9 | 1.9 | 2.3 | 2.1 | 1.4
  56 Days after 1st Vaccine: number analyzed (Participants) | 24 | 26 | 26 | 28 | 22 | 22 | 32 | 31
  56 Days after 1st Vaccine | 1.5 | 2.0 | 1.8 | 1.7 | 2.4 | 3.0 | 2.0 | 2.3
  168 Days after 1st Vaccine: number analyzed (Participants) | 24 | 25 | 26 | 25 | 22 | 21 | 31 | 31
  168 Days after 1st Vaccine | 1.8 | 4.3 | 1.8 | 1.0 | 1.1 | 0.2 | 2.9 | 3.6
  252 Days after 1st Vaccine: number analyzed (Participants) | 24 | 24 | 26 | 22 | 18 | 20 | 27 | 30
  252 Days after 1st Vaccine | 1.0 | 1.4 | 1.3 | 4.2 | 3.2 | 1.3 | 0.7 | 1.0
  365 Days after 1st Vaccine: number analyzed (Participants) | 22 | 23 | 26 | 23 | 18 | 20 | 27 | 30
  365 Days after 1st Vaccine | 0.4 | 0.9 | 0.9 | 0.9 | 1.2 | 1.0 | 0.7 | 0.9

5. Secondary Outcome: Relative Difference Expressed as a Percent in Vaccine-induced Antibodies to SARS-CoV-2 Antigens Over Time (S1-RBD IgA)
Description: Anti-S1-RBD protein. Relative difference is calculated as: [(LS Geometric Mean Active Arm - LS Geometric Mean Vaccine Alone Arm) / LS Geometric Mean Vaccine Alone Arm] x 100%
Time Frame: Up to 365 Days from 1st dose of Vaccination
Population: as for outcome 3
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 300 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 150 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 48 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 12 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 7 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 SC | REGN10933+REGN10987 + Vaccine 600 mg Day 1 SC
Number analyzed (Participants) | 26 | 26 | 26 | 28 | 24 | 24 | 32 | 32
Percent
  Baseline | -9.8 [-24.4 to 7.5] | -2.3 [-18.1 to 16.6] | -10.1 [-24.7 to 7.2] | 5.0 [-11.6 to 24.8] | 13.7 [-5.1 to 36.2] | 13.3 [-5.7 to 36.1] | 6.0 [-10.2 to 25.2] | -4.7 [-19.3 to 12.6]
  6 Days after 1st Vaccine: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 24 | 0 | 0
  6 Days after 1st Vaccine |  |  |  |  |  | -28.7 [-80.7 to 163.6] |  |
  14 Days after 1st Vaccine: number analyzed (Participants) | 26 | 25 | 25 | 28 | 24 | 24 | 31 | 32
  14 Days after 1st Vaccine | -15.3 [-54.4 to 57.1] | -6.2 [-49.9 to 75.5] | -43.6 [-69.9 to 5.5] | -31.6 [-62.6 to 25.2] | -33.9 [-64.9 to 24.7] | -35.0 [-65.5 to 22.7] | 5.2 [-41.5 to 89.2] | -3.2 [-46.1 to 73.7]
  28 Days after 1st Vaccine | -37.3 [-65.1 to 12.6] | -48.6 [-71.4 to -7.7] | -52.3 [-73.5 to -14.3] | -43.6 [-68.2 to -0.1] | -51.6 [-73.5 to -11.8] | -32.5 [-63.0 to 23.2] | -24.0 [-56.2 to 31.8] | -50.9 [-71.8 to -14.5]
  42 Days after 1st Vaccine: number analyzed (Participants) | 25 | 26 | 26 | 28 | 21 | 20 | 32 | 31
  42 Days after 1st Vaccine | -28.3 [-55.9 to 16.6] | -28.3 [-55.7 to 16.0] | -29.8 [-56.6 to 13.4] | -22.3 [-51.4 to 24.3] | -53.3 [-72.1 to -21.9] | -54.6 [-73.1 to -23.5] | -39.4 [-61.4 to -4.7] | -32.6 [-57.4 to 6.7]
  56 Days after 1st Vaccine: number analyzed (Participants) | 24 | 26 | 26 | 28 | 22 | 22 | 32 | 31
  56 Days after 1st Vaccine | -31.6 [-59.9 to 16.9] | -44.7 [-67.2 to -6.7] | -41.8 [-65.5 to -1.9] | -28.9 [-57.4 to 18.5] | -59.9 [-76.9 to -30.5] | -55.1 [-74.1 to -22.2] | -41.9 [-64.5 to -5.1] | -40.9 [-64.1 to -2.6]
  168 Days after 1st Vaccine: number analyzed (Participants) | 24 | 25 | 26 | 25 | 22 | 21 | 31 | 31
  168 Days after 1st Vaccine | -49.8 [-76.6 to 7.6] | -71.8 [-86.7 to -4.0] | -47.8 [-75.2 to 9.9] | 7.1 [-49.6 to 127.2] | -41.2 [-73.1 to 28.9] | 66.1 [-25.0 to 267.7] | -59.3 [-79.9 to -17.5] | -72.7 [-86.6 to -44.5]
  252 Days after 1st Vaccine: number analyzed (Participants) | 24 | 24 | 26 | 22 | 18 | 20 | 27 | 30
  252 Days after 1st Vaccine | -23.2 [-68.9 to 89.3] | -49.4 [-79.5 to 25.2] | -16.9 [-65.6 to 100.5] | -59.9 [-84.2 to 1.7] | -58.1 [-84.4 to 12.6] | -23.4 [-70.5 to 99.2] | 6.9 [-55.3 to 155.8] | -26.2 [-68.6 to 73.0]
  365 Days after 1st Vaccine: number analyzed (Participants) | 22 | 23 | 26 | 23 | 18 | 20 | 27 | 30
  365 Days after 1st Vaccine | 78.4 [-10.0 to 253.7] | 0.6 [-48.8 to 97.9] | 39.0 [-27.4 to 166.2] | 3.0 [-47.6 to 102.5] | -19.7 [-61.3 to 66.6] | 19.5 [-40.9 to 141.7] | 30.4 [-31.5 to 148.3] | 31.6 [-29.8 to 146.9]

6. Secondary Outcome: Absolute Values in Concentrations of Vaccine-induced Antibodies to SARS-CoV-2 Antigens Over Time (S-IgA)
Description: - Anti-S protein (Spike protein)
Time Frame: Up to 365 Days from 1st dose of Vaccination
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Binding Antibody Unit (BAU)/mL
Arm/Group | Vaccine Only | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 300 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 150 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 48 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 12 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 7 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 SC | REGN10933+REGN10987 + Vaccine 600 mg Day 1 SC
Number analyzed (Participants) | 42 | 26 | 26 | 26 | 28 | 24 | 24 | 32 | 32
Binding Antibody Unit (BAU)/mL
  Baseline: number analyzed (Participants) | 41 | 26 | 26 | 26 | 28 | 24 | 23 | 32 | 32
  Baseline | 11.7 (10.8) | 12.8 (15.7) | 8.5 (7.3) | 11.6 (14.7) | 14.2 (21.7) | 14.7 (26.1) | 17.3 (39.7) | 7.7 (3.8) | 12.9 (18.6)
  6 Days after 1st Vaccine: number analyzed (Participants) | 5 | 0 | 0 | 0 | 0 | 0 | 24 | 0 | 0
  6 Days after 1st Vaccine | 27.1 (29.2) |  |  |  |  |  | 662.5 (3155.1) |  |
  14 Days after 1st Vaccine: number analyzed (Participants) | 42 | 26 | 25 | 25 | 28 | 24 | 24 | 31 | 32
  14 Days after 1st Vaccine | 1597.4 (2367.2) | 1319.8 (1020.4) | 1984.7 (2708.3) | 1003.7 (1102.0) | 1020.7 (879.1) | 970.4 (1165.0) | 1636.9 (3070.8) | 1742.4 (2871.0) | 1494.4 (2303.0)
  28 Days after 1st Vaccine | 522.1 (466.7) | 400.1 (534.2) | 337.5 (386.9) | 246.6 (207.4) | 321.4 (309.2) | 343.1 (490.0) | 581.7 (1292.8) | 434.5 (425.0) | 349.0 (518.6)
  42 Days after 1st Vaccine: number analyzed (Participants) | 41 | 25 | 26 | 26 | 28 | 21 | 20 | 32 | 31
  42 Days after 1st Vaccine | 3147.1 (2905.2) | 2868.6 (2645.0) | 2472.4 (2243.8) | 2765.6 (3830.7) | 2396.0 (1923.4) | 1892.7 (1462.3) | 2089.8 (2548.4) | 2080.7 (1477.7) | 2029.1 (1652.4)
  56 Days after 1st Vaccine: number analyzed (Participants) | 41 | 24 | 26 | 26 | 28 | 22 | 22 | 32 | 31
  56 Days after 1st Vaccine | 1393.0 (1232.5) | 1218.0 (1192.6) | 941.5 (817.6) | 858.8 (849.3) | 1013.9 (818.1) | 813.1 (753.4) | 872.3 (1076.6) | 1009.6 (1182.4) | 911.9 (889.7)
  168 Days after 1st Vaccine: number analyzed (Participants) | 40 | 24 | 25 | 26 | 25 | 22 | 21 | 31 | 31
  168 Days after 1st Vaccine | 2060.3 (3446.9) | 931.9 (1466.0) | 405.6 (568.3) | 1378.0 (3168.9) | 1966.2 (3280.9) | 1251.0 (3206.3) | 2982.3 (3720.5) | 702.1 (1502.8) | 354.8 (591.3)
  252 Days after 1st Vaccine: number analyzed (Participants) | 37 | 24 | 24 | 26 | 22 | 18 | 20 | 27 | 30
  252 Days after 1st Vaccine | 4666.6 (5091.4) | 3753.9 (3919.0) | 3940.5 (5162.1) | 3497.8 (3891.3) | 1341.3 (1963.8) | 1911.1 (3022.5) | 2867.2 (3284.6) | 5957.8 (5727.3) | 5012.0 (5693.1)
  365 Days after 1st Vaccine: number analyzed (Participants) | 37 | 22 | 23 | 26 | 23 | 18 | 20 | 27 | 30
  365 Days after 1st Vaccine | 2808.8 (2971.8) | 3549.5 (2982.6) | 2703.2 (2444.5) | 2903.6 (3225.5) | 2302.4 (3101.0) | 3204.6 (4670.9) | 2944.1 (3850.8) | 3717.2 (4290.7) | 3648.0 (4074.5)

7. Secondary Outcome: Fold Change of Concentrations of Vaccine-induced Antibodies to SARS-CoV-2 Antigens Over Time (S-IgA)
Description: Anti-S protein Fold Change based on medians = (median value in vaccine only arm / median value in the active arm)
Time Frame: Up to 365 Days from 1st dose of vaccination
Population: as for outcome 3
Measure: Number; unit: Fold Change
Arm/Group | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 300 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 150 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 48 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 12 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 7 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 SC | REGN10933+REGN10987 + Vaccine 600 mg Day 1 SC
Number analyzed (Participants) | 26 | 26 | 26 | 28 | 24 | 24 | 32 | 32
Fold Change
  Baseline: number analyzed (Participants) | 26 | 26 | 26 | 28 | 24 | 23 | 32 | 32
  Baseline | 1.0 | 1.0 | 1.0 | 1.0 | 1.0 | 1.0 | 1.0 | 1.0
  6 Days after 1st Vaccine: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 24 | 0 | 0
  6 Days after 1st Vaccine |  |  |  |  |  | 0.7 |  |
  14 Days after 1st Vaccine: number analyzed (Participants) | 26 | 25 | 25 | 28 | 24 | 24 | 31 | 32
  14 Days after 1st Vaccine | 0.8 | 0.7 | 1.5 | 1.0 | 1.8 | 0.8 | 0.8 | 1.3
  28 Days after 1st Vaccine | 1.9 | 1.9 | 2.6 | 2.0 | 2.7 | 2.1 | 1.4 | 2.8
  42 Days after 1st Vaccine: number analyzed (Participants) | 25 | 26 | 26 | 28 | 21 | 20 | 32 | 31
  42 Days after 1st Vaccine | 1.4 | 1.6 | 1.7 | 1.6 | 1.5 | 1.5 | 1.7 | 1.9
  56 Days after 1st Vaccine: number analyzed (Participants) | 24 | 26 | 26 | 28 | 22 | 22 | 32 | 31
  56 Days after 1st Vaccine | 1.5 | 1.9 | 1.9 | 1.5 | 2.0 | 2.2 | 1.7 | 2.1
  168 Days after 1st Vaccine: number analyzed (Participants) | 24 | 25 | 26 | 25 | 22 | 21 | 31 | 31
  168 Days after 1st Vaccine | 1.5 | 2.2 | 1.6 | 0.9 | 1.1 | 0.2 | 1.6 | 2.6
  252 Days after 1st Vaccine: number analyzed (Participants) | 24 | 24 | 26 | 22 | 18 | 20 | 27 | 30
  252 Days after 1st Vaccine | 0.9 | 1.1 | 1.3 | 3.1 | 3.8 | 1.2 | 0.6 | 0.9
  365 Days after 1st Vaccine: number analyzed (Participants) | 22 | 23 | 26 | 23 | 18 | 20 | 27 | 30
  365 Days after 1st Vaccine | 0.6 | 1.0 | 1.0 | 1.0 | 1.1 | 1.3 | 0.8 | 1.0

8. Secondary Outcome: Relative Difference Expressed as a Percent in Vaccine-induced Antibodies to SARS-CoV-2 Antigens Over Time (S-IgA)
Description: Anti-S protein Relative difference is calculated as: [(LS Geometric Mean Active Arm - LS Geometric Mean Vaccine Alone Arm) / LS Geometric Mean Vaccine Alone Arm] x 100%
Time Frame: Up to 365 Days from 1st dose of Vaccination
Population: as for outcome 3
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 300 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 150 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 48 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 12 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 7 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 SC | REGN10933+REGN10987 + Vaccine 600 mg Day 1 SC
Number analyzed (Participants) | 26 | 26 | 26 | 28 | 24 | 24 | 32 | 32
Percent
  Baseline: number analyzed (Participants) | 26 | 26 | 26 | 28 | 24 | 23 | 32 | 32
  Baseline | 0.8 [-26.7 to 38.5] | -20.2 [-42.0 to 9.8] | -8.8 [-33.6 to 25.4] | 3.0 [-24.6 to 40.6] | -3.2 [-30.2 to 34.1] | 2.2 [-26.6 to 42.3] | -23.1 [-43.0 to 3.7] | -5.6 [-30.1 to 27.6]
  6 Days after 1st Vaccine: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 24 | 0 | 0
  6 Days after 1st Vaccine |  |  |  |  |  | -2.3 [-80.9 to 398.9] |  |
  14 Days after 1st Vaccine: number analyzed (Participants) | 26 | 25 | 25 | 28 | 24 | 24 | 31 | 32
  14 Days after 1st Vaccine | -3.7 [-43.7 to 64.7] | 1.8 [-40.9 to 75.5] | -34.7 [-62.1 to 12.5] | -22.9 [-54.4 to 30.4] | -27.4 [-58.2 to 25.9] | -21.6 [-54.8 to 36.1] | 10.4 [-33.7 to 83.8] | 8.8 [-34.6 to 80.7]
  28 Days after 1st Vaccine | -36.8 [-62.2 to 5.9] | -50.5 [-70.5 to -17.1] | -53.6 [-72.3 to -22.2] | -44.2 [-66.3 to -7.6] | -51.8 [-71.6 to -18.2] | -40.4 [-64.9 to 1.2] | -23.9 [-53.1 to 23.7] | -48.7 [-68.5 to -16.4]
  42 Days after 1st Vaccine: number analyzed (Participants) | 25 | 26 | 26 | 28 | 21 | 20 | 32 | 31
  42 Days after 1st Vaccine | -18.5 [-47.2 to 25.9] | -24.0 [-50.6 to 16.7] | -25.3 [-51.3 to 14.8] | -16.5 [-45.1 to 26.9] | -39.4 [-61.7 to -4.1] | -39.8 [-62.3 to -4.1] | -29.9 [-53.2 to 5.0] | -36.7 [-58.0 to -4.5]
  56 Days after 1st Vaccine: number analyzed (Participants) | 24 | 26 | 26 | 28 | 22 | 22 | 32 | 31
  56 Days after 1st Vaccine | -21.5 [-50.8 to 25.5] | -35.0 [-58.9 to 2.7] | -42.7 [-63.7 to -9.4] | -22.8 [-50.6 to 20.8] | -54.5 [-71.9 to -26.3] | -47.5 [-67.6 to -15.0] | -33.5 [-56.7 to 2.3] | -39.9 [-61.1 to -6.9]
  168 Days after 1st Vaccine: number analyzed (Participants) | 24 | 25 | 26 | 25 | 22 | 21 | 31 | 31
  168 Days after 1st Vaccine | -41.5 [-70.7 to 16.9] | -66.8 [-83.3 to -34.2] | -46.7 [-72.9 to 4.7] | 11.4 [-43.8 to 120.6] | -36.9 [-69.1 to 28.6] | 63.2 [-20.7 to 235.9] | -56.8 [-77.2 to -17.8] | -70.1 [-84.3 to -42.9]
  252 Days after 1st Vaccine: number analyzed (Participants) | 24 | 24 | 26 | 22 | 18 | 20 | 27 | 30
  252 Days after 1st Vaccine | -23.9 [-68.2 to 82.1] | -47.5 [-78.1 to 25.8] | -23.6 [-67.4 to 79.1] | -63.8 [-85.3 to -11.0] | -58.4 [-84.0 to 8.4] | -29.9 [-72.1 to 76.5] | 18.1 [-49.2 to 174.4] | -23.9 [-66.6 to 73.5]
  365 Days after 1st Vaccine: number analyzed (Participants) | 22 | 23 | 26 | 23 | 18 | 20 | 27 | 30
  365 Days after 1st Vaccine | 44.4 [-23.5 to 172.5] | 4.4 [-44.3 to 95.5] | 11.3 [-39.1 to 103.4] | -7.6 [-50.6 to 72.9] | -17.6 [-58.2 to 62.3] | -0.0 [-48.0 to 92.2] | 13.2 [-37.7 to 105.8] | 26.0 [-29.7 to 126.0]

9. Secondary Outcome: Absolute Values in Concentrations of Vaccine-induced Antibodies to SARS-CoV-2 Antigens Over Time (S-IgG)
Description: Anti-S protein
Time Frame: Up to 365 Days from 1st dose of vaccination
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Binding Antibody Unit (BAU)/mL
Arm/Group | Vaccine Only | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 300 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 150 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 48 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 12 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 7 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 SC | REGN10933+REGN10987 + Vaccine 600 mg Day 1 SC
Number analyzed (Participants) | 42 | 26 | 26 | 26 | 28 | 24 | 24 | 32 | 32
Binding Antibody Unit (BAU)/mL
  Baseline: number analyzed (Participants) | 41 | 26 | 26 | 26 | 28 | 24 | 23 | 30 | 26
  Baseline | 4.5 (3.9) | 8.1 (10.4) | 4.4 (2.7) | 3.2 (1.2) | 5.9 (6.7) | 59.8 (267.1) | 5.1 (5.4) | 3.0 (1.4) | 4.0 (3.3)
  6 Days after 1st Vaccine: number analyzed (Participants) | 5 | 0 | 0 | 0 | 0 | 0 | 24 | 0 | 0
  6 Days after 1st Vaccine | 4.0 (1.8) |  |  |  |  |  | 624.8 (3025.9) |  |
  14 Days after 1st Vaccine: number analyzed (Participants) | 42 | 26 | 25 | 25 | 28 | 24 | 24 | 31 | 32
  14 Days after 1st Vaccine | 409.7 (527.4) | 600.2 (1399.6) | 205.9 (175.8) | 256.3 (298.9) | 1742.9 (5319.5) | 497.1 (1620.0) | 1059.4 (3414.4) | 211.8 (226.6) | 345.1 (679.0)
  28 Days after 1st Vaccine | 676.8 (878.5) | 468.6 (860.3) | 173.3 (137.1) | 183.7 (168.5) | 1450.6 (4361.4) | 366.7 (1040.5) | 973.5 (3309.8) | 318.2 (390.6) | 598.7 (2096.6)
  42 Days after 1st Vaccine: number analyzed (Participants) | 41 | 25 | 26 | 26 | 28 | 21 | 20 | 32 | 31
  42 Days after 1st Vaccine | 4900.0 (3970.8) | 3814.3 (3083.2) | 2769.7 (2535.4) | 2816.7 (2858.9) | 5074.9 (6044.3) | 2179.8 (928.5) | 3968.7 (3806.8) | 2797.7 (1787.2) | 2852.9 (2450.6)
  56 Days after 1st Vaccine: number analyzed (Participants) | 41 | 24 | 26 | 26 | 28 | 22 | 22 | 32 | 31
  56 Days after 1st Vaccine | 3459.1 (3498.4) | 3737.3 (4638.6) | 1841.8 (1012.7) | 1849.9 (1693.2) | 3432.9 (5246.8) | 2227.5 (2300.0) | 3358.0 (4515.3) | 1980.6 (1470.2) | 2361.7 (2513.4)
  168 Days after 1st Vaccine: number analyzed (Participants) | 40 | 24 | 25 | 26 | 25 | 22 | 21 | 31 | 31
  168 Days after 1st Vaccine | 2208.7 (3093.8) | 2156.7 (4354.7) | 900.0 (2018.7) | 1862.8 (3723.4) | 2973.3 (4045.5) | 1346.4 (1762.0) | 4609.3 (5678.3) | 940.1 (1486.8) | 729.5 (889.1)
  252 Days after 1st Vaccine: number analyzed (Participants) | 37 | 24 | 24 | 26 | 22 | 18 | 20 | 27 | 30
  252 Days after 1st Vaccine | 6319.0 (6625.5) | 5682.5 (6074.3) | 4138.0 (5343.0) | 7004.3 (7077.5) | 4784.2 (4832.5) | 4974.1 (6150.0) | 6830.1 (5394.9) | 6806.3 (7138.7) | 6855.6 (7833.3)
  365 Days after 1st Vaccine: number analyzed (Participants) | 37 | 22 | 23 | 26 | 23 | 18 | 20 | 27 | 30
  365 Days after 1st Vaccine | 5724.1 (4944.5) | 8865.1 (7110.6) | 7888.9 (7014.8) | 7596.9 (7438.6) | 4954.4 (5226.5) | 5263.3 (6235.8) | 3819.3 (3262.7) | 9836.6 (7299.8) | 10863.1 (7822.4)

10. Secondary Outcome: Fold Change of Concentrations of Vaccine-induced Antibodies to SARS-CoV-2 Antigens Over Time (S-IgG)
Description: Anti-S protein Fold Change based on medians = (median value in vaccine only arm / median value in the active arm)
Time Frame: Up to 365 Days from 1st dose of vaccination
Population: as for outcome 3
Measure: Number; unit: Fold Change
Arm/Group | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 300 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 150 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 48 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 12 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 7 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 SC | REGN10933+REGN10987 + Vaccine 600 mg Day 1 SC
Number analyzed (Participants) | 26 | 26 | 26 | 28 | 24 | 24 | 32 | 32
Fold Change
  Baseline: number analyzed (Participants) | 26 | 26 | 26 | 28 | 24 | 23 | 32 | 32
  Baseline | 0.4 | 1.0 | 1.0 | 1.0 | 1.0 | 1.0 | 1.0 | 1.0
  6 Days after 1st Vaccine: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 24 | 0 | 0
  6 Days after 1st Vaccine |  |  |  |  |  | 0.5 |  |
  14 Days after 1st Vaccine: number analyzed (Participants) | 26 | 25 | 25 | 28 | 24 | 24 | 31 | 32
  14 Days after 1st Vaccine | 1.6 | 1.7 | 1.8 | 3.5 | 2.5 | 1.0 | 2.4 | 2.1
  28 Days after 1st Vaccine | 3.1 | 4.1 | 3.7 | 2.8 | 3.7 | 2.6 | 2.3 | 2.9
  42 Days after 1st Vaccine: number analyzed (Participants) | 25 | 26 | 26 | 28 | 21 | 20 | 32 | 31
  42 Days after 1st Vaccine | 1.1 | 1.5 | 1.6 | 1.1 | 1.4 | 1.2 | 1.3 | 1.4
  56 Days after 1st Vaccine: number analyzed (Participants) | 24 | 26 | 26 | 28 | 22 | 22 | 32 | 31
  56 Days after 1st Vaccine | 1.2 | 1.5 | 1.8 | 1.1 | 1.4 | 1.6 | 1.6 | 1.6
  168 Days after 1st Vaccine: number analyzed (Participants) | 24 | 25 | 26 | 25 | 22 | 21 | 31 | 31
  168 Days after 1st Vaccine | 1.7 | 1.7 | 1.8 | 0.4 | 1.1 | 0.4 | 1.3 | 1.5
  252 Days after 1st Vaccine: number analyzed (Participants) | 24 | 24 | 26 | 22 | 18 | 20 | 27 | 30
  252 Days after 1st Vaccine | 1.1 | 1.4 | 0.6 | 1.2 | 1.2 | 0.5 | 1.0 | 1.2
  365 Days after 1st Vaccine: number analyzed (Participants) | 22 | 23 | 26 | 23 | 18 | 20 | 27 | 30
  365 Days after 1st Vaccine | 0.7 | 0.7 | 0.9 | 1.6 | 1.8 | 1.4 | 0.5 | 0.5

11. Secondary Outcome: Relative Difference Expressed as a Percent in Vaccine-induced Antibodies to SARS-CoV-2 Antigens Over Time (S-IgG)
Description: Anti-S protein (Spike) Relative difference is calculated as: [(LS Geometric Mean Active Arm - LS Geometric Mean Vaccine Alone Arm) / LS Geometric Mean Vaccine Alone Arm] x 100%
Time Frame: Up to 365 Days from 1st dose of vaccination
Population: as for outcome 3
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 300 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 150 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 48 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 12 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 7 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 SC | REGN10933+REGN10987 + Vaccine 600 mg Day 1 SC
Number analyzed (Participants) | 26 | 26 | 26 | 28 | 24 | 24 | 32 | 32
Percent
  Baseline: number analyzed (Participants) | 26 | 26 | 26 | 28 | 24 | 23 | 32 | 32
  Baseline | 58.9 [15.4 to 118.9] | 3.0 [-25.3 to 41.9] | -18.7 [-41.0 to 12.0] | 18.3 [-13.5 to 61.9] | 29.4 [-6.9 to 79.8] | 5.4 [-24.5 to 47.1] | -22.9 [-43.0 to 4.2] | -10.3 [-33.8 to 21.5]
  6 Days after 1st Vaccine: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 24 | 0 | 0
  6 Days after 1st Vaccine |  |  |  |  |  | 88.0 [-65.3 to 919.3] |  |
  14 Days after 1st Vaccine: number analyzed (Participants) | 26 | 26 | 25 | 25 | 24 | 24 | 31 | 32
  14 Days after 1st Vaccine | -25.1 [-60.2 to 41.0] | -48.5 [-72.9 to -2.1] | -44.5 [-70.8 to 5.4] | -29.9 [-62.2 to 30.2] | -47.8 [-72.8 to -0.2] | 8.2 [-43.5 to 107.0] | -34.0 [-63.8 to 20.3] | -28.3 [-60.6 to 30.4]
  28 Days after 1st Vaccine: number analyzed (Participants) | 26 | 25 | 26 | 26 | 24 | 24 | 32 | 32
  28 Days after 1st Vaccine | -45.5 [-70.6 to 1.0] | -64.1 [-80.6 to -33.4] | -63.4 [-80.3 to -32.1] | -33.8 [-63.8 to 21.0] | -57.0 [-77.2 to -19.1] | -28.4 [-62.0 to 34.9] | -38.6 [-65.6 to 9.8] | -45.7 [-69.7 to -2.6]
  42 Days after 1st Vaccine: number analyzed (Participants) | 25 | 26 | 26 | 28 | 21 | 20 | 32 | 31
  42 Days after 1st Vaccine | -25.5 [-52.2 to 16.3] | -50.1 [-67.9 to -22.6] | -45.9 [-65.1 to -16.0] | -15.3 [-44.9 to 30.2] | -46.7 [-66.7 to -14.7] | -46.4 [-66.8 to -13.5] | -35.4 [-57.3 to -2.3] | -34.7 [-57.1 to -0.6]
  56 Days after 1st Vaccine: number analyzed (Participants) | 24 | 26 | 26 | 28 | 22 | 22 | 32 | 31
  56 Days after 1st Vaccine | 6.2 [-33.3 to 69.1] | -34.8 [-58.6 to 2.8] | -36.6 [-59.7 to -0.1] | -6.9 [-40.3 to 45.1] | -23.6 [-52.7 to 23.3] | -18.9 [-49.8 to 30.9] | -29.1 [-53.8 to 8.7] | -20.9 [-48.8 to 22.1]
  168 Days after 1st Vaccine: number analyzed (Participants) | 24 | 25 | 26 | 25 | 22 | 21 | 31 | 31
  168 Days after 1st Vaccine | -29.1 [-61.4 to 30.1] | -54.2 [-74.9 to -16.5] | -29.5 [-61.0 to 27.5] | 48.6 [-18.4 to 170.8] | -9.3 [-51.5 to 69.4] | 98.9 [5.6 to 274.8] | -40.6 [-66.2 to 4.3] | -48.0 [-70.5 to -8.3]
  252 Days after 1st Vaccine: number analyzed (Participants) | 24 | 24 | 26 | 22 | 18 | 20 | 27 | 30
  252 Days after 1st Vaccine | -13.4 [-61.3 to 93.9] | -47.4 [-76.6 to 17.9] | 4.4 [-52.4 to 129.3] | -2.6 [-57.6 to 123.5] | -5.2 [-60.8 to 129.3] | 49.1 [-36.4 to 249.7] | 28.2 [-41.2 to 179.4] | -12.2 [-59.0 to 87.9]
  365 Days after 1st Vaccine: number analyzed (Participants) | 22 | 23 | 26 | 23 | 18 | 20 | 27 | 30
  365 Days after 1st Vaccine | 65.6 [-10.0 to 204.6] | 44.0 [-21.1 to 163.0] | 38.1 [-22.6 to 146.4] | -3.1 [-46.9 to 76.9] | -20.2 [-58.3 to 53.0] | -23.9 [-59.4 to 42.4] | 78.7 [0.7 to 217.0] | 116.6 [23.7 to 279.3]

12. Secondary Outcome: Absolute Values in Concentrations of Vaccine-induced Antibodies to SARS-CoV-2 Antigens Over Time (S1-RBD IgG)
Description: Anti-S1-RBD
Time Frame: Up to 365 Days from 1st dose of vaccination
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Binding Antibody Unit (BAU)/mL
Arm/Group | Vaccine Only | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 300 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 150 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 48 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 12 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 7 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 SC | REGN10933+REGN10987 + Vaccine 600 mg Day 1 SC
Number analyzed (Participants) | 42 | 26 | 26 | 26 | 28 | 24 | 24 | 32 | 32
Binding Antibody Unit (BAU)/mL
  Baseline: number analyzed (Participants) | 41 | 26 | 26 | 26 | 28 | 24 | 23 | 32 | 32
  Baseline | 6.6 (4.0) | 14.0 (21.4) | 6.8 (2.8) | 5.6 (3.0) | 9.0 (6.0) | 111.4 (512.7) | 9.2 (8.7) | 5.4 (2.4) | 7.5 (10.3)
  6 Days after 1st Vaccine: number analyzed (Participants) | 5 | 0 | 0 | 0 | 0 | 0 | 24 | 0 | 0
  6 Days after 1st Vaccine | 7.2 (2.8) |  |  |  |  |  | 940.8 (4569.2) |  |
  14 Days after 1st Vaccine: number analyzed (Participants) | 42 | 26 | 25 | 25 | 28 | 24 | 24 | 31 | 32
  14 Days after 1st Vaccine | 403.4 (650.2) | 521.4 (1411.9) | 185.9 (262.0) | 153.1 (218.2) | 2830.5 (9711.1) | 493.7 (1936.3) | 1340.3 (5510.0) | 159.7 (165.2) | 290.9 (729.9)
  28 Days after 1st Vaccine | 809.4 (1100.8) | 448.4 (841.7) | 206.0 (177.2) | 182.3 (214.1) | 2050.2 (6594.9) | 418.5 (1282.0) | 1417.6 (5411.7) | 353.5 (434.6) | 597.0 (2153.3)
  42 Days after 1st Vaccine: number analyzed (Participants) | 41 | 25 | 26 | 26 | 28 | 21 | 20 | 32 | 31
  42 Days after 1st Vaccine | 7638.6 (7214.2) | 7336.3 (6920.7) | 4969.6 (4706.1) | 4776.7 (5241.9) | 10764.3 (17718.4) | 3229.9 (1467.4) | 5665.7 (5297.2) | 4342.8 (3047.2) | 4537.6 (4153.6)
  56 Days after 1st Vaccine: number analyzed (Participants) | 41 | 24 | 26 | 26 | 28 | 22 | 22 | 32 | 31
  56 Days after 1st Vaccine | 5595.6 (6439.6) | 6945.4 (10762.4) | 3123.9 (1915.7) | 3148.8 (3404.7) | 7023.8 (14395.7) | 4077.9 (4581.2) | 4864.7 (6282.4) | 3080.5 (2507.4) | 3775.4 (3840.3)
  168 Days after 1st Vaccine: number analyzed (Participants) | 40 | 24 | 25 | 26 | 25 | 22 | 21 | 31 | 31
  168 Days after 1st Vaccine | 4007.7 (6218.6) | 4208.6 (9593.8) | 1578.5 (3810.3) | 3438.9 (7459.7) | 5873.1 (9336.1) | 2243.6 (3035.3) | 10359.9 (14463.6) | 1372.4 (2310.7) | 1262.8 (1957.9)
  252 Days after 1st Vaccine: number analyzed (Participants) | 37 | 24 | 24 | 26 | 22 | 18 | 20 | 27 | 30
  252 Days after 1st Vaccine | 13505.1 (15811.0) | 13428.1 (15027.8) | 9549.2 (14673.8) | 1487.0 (18618.2) | 9124.4 (11583.7) | 11189.1 (16641.6) | 12902.6 (10578.8) | 14503.6 (19241.8) | 17456.8 (23681.5)
  365 Days after 1st Vaccine: number analyzed (Participants) | 37 | 22 | 23 | 26 | 23 | 18 | 20 | 27 | 30
  365 Days after 1st Vaccine | 11268.3 (11087.5) | 21517.0 (23659.3) | 16569.7 (15884.0) | 16959.2 (20989.3) | 10225.9 (13257.7) | 11261.7 (15375.7) | 6301.3 (5284.8) | 19774.5 (16462.8) | 23135.5 (19481.4)

13. Secondary Outcome: Fold Change of Concentrations of Vaccine-induced Antibodies to SARS-CoV-2 Antigens Over Time (S1-RBD IgG)
Description: Anti-S1-RBD protein Fold Change based on medians = (median value in vaccine only arm / median value in the active arm)
Time Frame: Up to 365 Days from 1st dose of vaccination
Population: as for outcome 3
Measure: Number; unit: Fold Change
Arm/Group | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 300 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 150 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 48 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 12 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 7 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 SC | REGN10933+REGN10987 + Vaccine 600 mg Day 1 SC
Number analyzed (Participants) | 26 | 26 | 26 | 28 | 24 | 24 | 32 | 32
Fold Change
  Baseline: number analyzed (Participants) | 26 | 26 | 26 | 28 | 24 | 23 | 32 | 32
  Baseline | 0.4 | 0.7 | 1.0 | 0.5 | 1.0 | 1.0 | 1.0 | 1.0
  6 Days after 1st Vaccine: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 24 | 0 | 0
  6 Days after 1st Vaccine |  |  |  |  |  | 1.0 |  |
  14 Days after 1st Vaccine: number analyzed (Participants) | 26 | 25 | 25 | 28 | 24 | 24 | 31 | 32
  14 Days after 1st Vaccine | 2.1 | 2.3 | 3.4 | 3.5 | 3.0 | 1.3 | 2.3 | 2.6
  28 Days after 1st Vaccine | 2.8 | 3.5 | 4.2 | 2.6 | 4.0 | 2.2 | 2.2 | 2.7
  42 Days after 1st Vaccine: number analyzed (Participants) | 25 | 26 | 26 | 28 | 21 | 20 | 32 | 31
  42 Days after 1st Vaccine | 1.1 | 1.3 | 1.5 | 1.0 | 1.4 | 1.3 | 1.3 | 1.2
  56 Days after 1st Vaccine: number analyzed (Participants) | 24 | 26 | 26 | 28 | 22 | 22 | 32 | 31
  56 Days after 1st Vaccine | 1.1 | 1.3 | 1.8 | 1.2 | 1.3 | 1.5 | 1.5 | 1.6
  168 Days after 1st Vaccine: number analyzed (Participants) | 24 | 25 | 26 | 25 | 22 | 21 | 31 | 31
  168 Days after 1st Vaccine | 1.8 | 1.6 | 1.5 | 0.4 | 0.9 | 0.3 | 1.3 | 1.5
  252 Days after 1st Vaccine: number analyzed (Participants) | 24 | 24 | 26 | 22 | 18 | 20 | 27 | 30
  252 Days after 1st Vaccine | 0.9 | 1.9 | 0.9 | 1.5 | 1.8 | 0.7 | 1.1 | 1.5
  365 Days after 1st Vaccine: number analyzed (Participants) | 22 | 23 | 26 | 23 | 18 | 20 | 27 | 30
  365 Days after 1st Vaccine | 0.7 | 0.6 | 0.8 | 1.4 | 1.6 | 1.4 | 0.5 | 0.4

14. Secondary Outcome: Relative Difference Expressed as a Percent in Vaccine-induced Antibodies to SARS-CoV-2 Antigens Over Time (S1-RBD IgG)
Description: Anti-S1-RBD protein Relative difference is calculated as: [(LS Geometric Mean Active Arm - LS Geometric Mean Vaccine Alone Arm) / LS Geometric Mean Vaccine Alone Arm] x 100%
Time Frame: Up to 365 Days from 1st dose of vaccination
Population: as for outcome 3
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 300 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 150 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 48 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 12 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 7 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 SC | REGN10933+REGN10987 + Vaccine 600 mg Day 1 SC
Number analyzed (Participants) | 26 | 26 | 26 | 28 | 24 | 24 | 32 | 32
Percent
  Baseline | 58.3 [13.8 to 120.2] | 7.3 [-22.9 to 49.4] | -13.0 [-37.5 to 21.1] | 27.5 [-7.7 to 76.1] | 25.8 [-10.4 to 76.5] | 18.2 [-16.2 to 66.7] | -14.3 [-37.2 to 17.0] | -9.0 [-33.4 to 24.4]
  6 Days after 1st Vaccine: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 24 | 0 | 0
  6 Days after 1st Vaccine |  |  |  |  |  | 43.3 [-72.8 to 654.8] |  |
  14 Days after 1st Vaccine: number analyzed (Participants) | 26 | 25 | 25 | 28 | 24 | 24 | 31 | 32
  14 Days after 1st Vaccine | -35.5 [-67.0 to 26.1] | -53.3 [-76.3 to -7.7] | -59.9 [-79.7 to -20.9] | -38.5 [-68.1 to 18.4] | -56.2 [-78.0 to -12.9] | -16.4 [-58.0 to 66.5] | -44.1 [-70.4 to 5.6] | -39.1 [-67.7 to 14.8]
  28 Days after 1st Vaccine | -50.8 [-74.3 to -6.0] | -66.0 [-82.2 to -34.8] | -71.3 [-85.0 to -45.0] | -43.2 [-69.8 to 7.1] | -60.6 [-79.7 to -23.4] | -40.7 [-69.5 to 15.2] | -46.4 [-70.9 to -1.5] | -52.0 [-74.0 to -11.5]
  42 Days after 1st Vaccine: number analyzed (Participants) | 25 | 26 | 26 | 28 | 21 | 20 | 32 | 31
  42 Days after 1st Vaccine | -11.8 [-45.9 to 43.7] | -41.2 [-63.7 to -4.6] | -40.7 [-63.4 to -3.8] | -0.0 [-37.6 to 60.3] | -44.0 [-66.6 to -6.1] | -46.4 [-68.3 to -9.4] | -30.3 [-55.8 to 9.8] | -27.5 [-54.3 to 15.1]
  56 Days after 1st Vaccine: number analyzed (Participants) | 24 | 26 | 26 | 28 | 22 | 22 | 32 | 31
  56 Days after 1st Vaccine | 14.8 [-29.8 to 87.5] | -29.3 [-56.2 to 14.2] | -34.5 [-59.4 to 5.8] | -0.3 [-37.6 to 59.2] | -10.8 [-46.2 to 47.8] | -19.1 [-51.2 to 34.1] | -28.3 [-54.4 to 12.5] | -14.2 [-45.7 to 35.6]
  168 Days after 1st Vaccine: number analyzed (Participants) | 24 | 25 | 26 | 25 | 22 | 21 | 31 | 31
  168 Days after 1st Vaccine | -26.0 [-62.0 to 44.1] | -50.5 [-74.4 to -4.3] | -20.4 [-58.4 to 52.6] | 60.7 [-16.8 to 210.5] | -3.1 [-51.2 to 92.5] | 135.3 [17.4 to 371.6] | -45.2 [-70.4 to 1.8] | -45.2 [-70.6 to 2.1]
  252 Days after 1st Vaccine: number analyzed (Participants) | 24 | 24 | 26 | 22 | 18 | 20 | 27 | 30
  252 Days after 1st Vaccine | -3.9 [-61.0 to 136.6] | -48.3 [-79.1 to 27.6] | 10.5 [-54.2 to 166.3] | -6.6 [-63.1 to 136.6] | -1.4 [-63.3 to 164.8] | 48.4 [-42.8 to 285.2] | 19.1 [-50.2 to 184.7] | 1.8 [-56.5 to 138.4]
  365 Days after 1st Vaccine: number analyzed (Participants) | 22 | 23 | 26 | 23 | 18 | 20 | 27 | 30
  365 Days after 1st Vaccine | 102.8 [4.5 to 293.4] | 63.5 [-15.1 to 214.7] | 45.5 [-22.5 to 173.1] | 2.7 [-46.6 to 97.5] | -14.9 [-58.1 to 72.6] | -27.8 [-63.5 to 42.8] | 82.8 [-2.0 to 241.1] | 145.7 [33.6 to 351.9]

15. Secondary Outcome: Absolute Values in Concentrations of Vaccine-induced Antibodies to SARS-CoV-2 Antigens Over Time (S1-RBD IgM)
Description: Anti-S1-RBD
Time Frame: Up to 365 Days from 1st dose of vaccination
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Binding Antibody Unit (BAU)/mL
Arm/Group | Vaccine Only | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 300 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 150 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 48 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 12 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 7 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 SC | REGN10933+REGN10987 + Vaccine 600 mg Day 1 SC
Number analyzed (Participants) | 42 | 26 | 26 | 26 | 28 | 24 | 24 | 32 | 32
Binding Antibody Unit (BAU)/mL
  Baseline: number analyzed (Participants) | 41 | 26 | 26 | 26 | 28 | 24 | 23 | 32 | 32
  Baseline | 7.0 (7.3) | 7.1 (5.2) | 7.5 (7.7) | 6.4 (4.1) | 6.5 (6.8) | 6.9 (4.2) | 7.0 (4.9) | 6.1 (3.2) | 5.7 (2.6)
  6 Days after 1st Vaccine: number analyzed (Participants) | 5 | 0 | 0 | 0 | 0 | 0 | 24 | 0 | 0
  6 Days after 1st Vaccine | 8.9 (6.8) |  |  |  |  |  | 13.1 (20.9) |  |
  14 Days after 1st Vaccine: number analyzed (Participants) | 42 | 26 | 25 | 25 | 28 | 24 | 24 | 31 | 32
  14 Days after 1st Vaccine | 53.8 (70.8) | 29.2 (38.7) | 25.5 (26.2) | 35.1 (64.5) | 852.6 (4399.3) | 14.3 (13.9) | 42.3 (47.9) | 774.5 (4180.7) | 34.4 (81.2)
  28 Days after 1st Vaccine | 34.5 (32.4) | 17.3 (22.3) | 14.8 (16.0) | 17.5 (25.1) | 848.9 (4400.0) | 14.2 (16.1) | 27.3 (28.1) | 750.8 (4114.9) | 17.9 (39.7)
  42 Days after 1st Vaccine: number analyzed (Participants) | 41 | 25 | 26 | 26 | 28 | 21 | 20 | 32 | 31
  42 Days after 1st Vaccine | 55.5 (57.2) | 38.5 (55.9) | 20.3 (16.8) | 21.7 (18.3) | 869.2 (4396.1) | 37.9 (33.7) | 40.5 (38.4) | 762.2 (4113.0) | 29.0 (35.5)
  56 Days after 1st Vaccine: number analyzed (Participants) | 41 | 24 | 26 | 26 | 28 | 22 | 22 | 32 | 31
  56 Days after 1st Vaccine | 34.1 (34.9) | 20.6 (29.4) | 11.8 (9.7) | 12.2 (9.3) | 37.0 (79.2) | 19.8 (16.7) | 27.1 (23.3) | 30.9 (63.0) | 17.6 (19.9)
  168 Days after 1st Vaccine: number analyzed (Participants) | 40 | 24 | 25 | 26 | 25 | 22 | 21 | 31 | 31
  168 Days after 1st Vaccine | 11.7 (9.5) | 8.9 (6.1) | 8.7 (10.6) | 10.8 (14.4) | 15.8 (22.1) | 9.4 (10.9) | 12.1 (9.2) | 9.1 (11.4) | 6.5 (4.4)
  252 Days after 1st Vaccine: number analyzed (Participants) | 37 | 24 | 24 | 26 | 22 | 18 | 20 | 27 | 30
  252 Days after 1st Vaccine | 13.6 (13.3) | 10.2 (6.9) | 11.1 (12.7) | 10.5 (9.1) | 17.9 (36.1) | 10.2 (12.6) | 12.8 (18.5) | 875.0 (4481.7) | 16.9 (22.8)
  365 Days after 1st Vaccine: number analyzed (Participants) | 37 | 22 | 23 | 26 | 23 | 18 | 20 | 27 | 30
  365 Days after 1st Vaccine | 9.2 (6.5) | 8.6 (5.6) | 8.1 (6.4) | 9.6 (9.7) | 13.7 (18.3) | 7.2 (5.7) | 14.6 (22.8) | 10.6 (15.7) | 11.8 (13.5)

16. Secondary Outcome: Relative Difference Expressed as a Percent in Vaccine-induced Antibodies to SARS-CoV-2 Antigens Over Time (S1-RBD IgM)
Description: as for outcome 14
Time Frame: Up to 365 Days from 1st dose of vaccination
Population: as for outcome 1
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 300 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 150 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 48 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 12 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 7 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 SC | REGN10933+REGN10987 + Vaccine 600 mg Day 1 SC
Number analyzed (Participants) | 26 | 26 | 26 | 28 | 24 | 24 | 32 | 32
Percent
  Baseline: number analyzed (Participants) | 26 | 26 | 26 | 28 | 24 | 23 | 32 | 32
  Baseline | 5.9 [-15.9 to 33.5] | 3.5 [-17.9 to 30.5] | -1.5 [-21.8 to 24.2] | -4.7 [-24.1 to 19.5] | 6.0 [-16.4 to 34.5] | 3.6 [-18.6 to 31.8] | -1.7 [-20.9 to 22.3] | -4.9 [-23.6 to 18.4]
  6 Days after 1st Vaccine: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  14 Days after 1st Vaccine: number analyzed (Participants) | 26 | 25 | 25 | 28 | 24 | 24 | 31 | 32
  14 Days after 1st Vaccine | -43.7 [-69.0 to 2.3] | -50.9 [-73.2 to -10.0] | -54.7 [-75.3 to -16.9] | -36.7 [-64.7 to 13.7] | -62.8 [-79.9 to -31.3] | -10.9 [-51.7 to 64.7] | -34.9 [-63.1 to 14.8] | -41.0 [-66.5 to 3.8]
  28 Days after 1st Vaccine | -46.6 [-70.0 to -5.1] | -53.6 [-73.9 to -17.3] | -53.3 [-73.8 to -17.0] | -26.5 [-58.2 to 29.0] | -52.0 [-73. to -13.4] | -15.5 [-53.2 to 52.5] | -27.7 [-57.9 to 24.3] | -51.3 [-71.7 to -16.0]
  42 Days after 1st Vaccine: number analyzed (Participants) | 25 | 26 | 26 | 28 | 21 | 20 | 32 | 31
  42 Days after 1st Vaccine | -22.7 [-56.1 to 36.4] | -55.9 [-74.8 to -22.7] | -51.5 [-72.3 to -15.1] | 8.0 [-37.6 to 86.8] | -18.2 [-55.1 to 49.2] | -20.2 [-56.6 to 46.9] | -36.3 [-62.4 to 8.0] | -43.0 [-66.7 to -2.5]
  56 Days after 1st Vaccine: number analyzed (Participants) | 24 | 26 | 26 | 28 | 22 | 22 | 32 | 31
  56 Days after 1st Vaccine | -33.6 [-58.8 to 7.2] | -58.2 [-73.8 to -33.2] | -56.6 [-72.8 to -30.8] | -16.8 [-47.3 to 31.3] | -32.9 [-59.0 to 9.8] | -14.0 [-47.5 to 40.6] | -37.7 [-59.8 to -3.2] | -42.3 [-63.1 to -9.8]
  168 Days after 1st Vaccine: number analyzed (Participants) | 24 | 25 | 26 | 25 | 22 | 21 | 31 | 31
  168 Days after 1st Vaccine | -18.5 [-42.5 to 15.5] | -30.5 [-50.8 to -1.8] | -17.8 [-41.5 to 15.6] | 6.8 [-24.3 to 50.8] | -23.8 [-46.8 to 9.1] | 3.2 [-28.3 to 48.5] | -27.3 [-47.4 to 0.5] | -35.4 [-53.4 to -10.5]
  252 Days after 1st Vaccine: number analyzed (Participants) | 24 | 24 | 26 | 22 | 18 | 20 | 27 | 30
  252 Days after 1st Vaccine | -15.2 [-48.4 to 39.1] | -20.0 [-51.3 to 31.6] | -19.3 [-50.3 to 30.9] | -17.2 [-50.3 to 38.1] | -22.3 [-54.9 to 33.8] | -13.0 [-48.5 to 46.9] | 20.6 [-25.3 to 94.8] | 6.4 [-33.4 to 69.9]
  365 Days after 1st Vaccine: number analyzed (Participants) | 22 | 23 | 26 | 23 | 18 | 20 | 27 | 30
  365 Days after 1st Vaccine | -4.0 [-34.7 to 41.1] | -12.4 [-40.2 to 28.1] | -6.6 [-35.2 to 34.7] | 8.3 [-26.0 to 58.4] | -19.1 [-46.4 to 22.1] | 13.5 [-23.7 to 68.8] | -8.7 [-36.5 to 31.2] | 8.1 [-24.1 to 54.1]

17. Secondary Outcome: Fold Change of Concentrations of Vaccine-induced Antibodies to SARS-CoV-2 Antigens Over Time (S1-RBD IgM)
Description: Anti-S1-RBD protein Fold Change based on medians = (median value in vaccine only arm / median value in the active arm)
Time Frame: Up to 365 Days from 1st dose of vaccination
Population: as for outcome 1
Measure: Number; unit: Fold Change
Arm/Group | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 300 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 150 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 48 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 12 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 7 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 SC | REGN10933+REGN10987 + Vaccine 600 mg Day 1 SC
Number analyzed (Participants) | 26 | 26 | 26 | 28 | 24 | 24 | 32 | 32
Fold Change
  Baseline | 1.0 | 1.0 | 1.0 | 1.0 | 1.0 | 1.0 | 1.0 | 1.0
  6 Days after 1st Vaccine: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  14 Days after 1st Vaccine: number analyzed (Participants) | 26 | 25 | 25 | 28 | 24 | 24 | 31 | 32
  14 Days after 1st Vaccine | 1.9 | 1.8 | 2.6 | 2.4 | 3.3 | 1.0 | 2.1 | 2.3
  28 Days after 1st Vaccine | 2.3 | 3.1 | 5.0 | 2.1 | 5.0 | 1.4 | 2.3 | 5.0
  42 Days after 1st Vaccine: number analyzed (Participants) | 25 | 26 | 26 | 28 | 21 | 20 | 32 | 31
  42 Days after 1st Vaccine | 2.0 | 2.4 | 2.8 | 1.6 | 1.9 | 1.5 | 3.1 | 2.3
  56 Days after 1st Vaccine: number analyzed (Participants) | 24 | 26 | 26 | 28 | 22 | 22 | 32 | 31
  56 Days after 1st Vaccine | 1.5 | 2.8 | 2.8 | 1.1 | 1.4 | 0.9 | 1.7 | 1.6
  168 Days after 1st Vaccine: number analyzed (Participants) | 24 | 25 | 26 | 25 | 22 | 21 | 31 | 31
  168 Days after 1st Vaccine | 2.1 | 2.1 | 2.1 | 2.1 | 2.1 | 0.9 | 2.1 | 2.1
  252 Days after 1st Vaccine: number analyzed (Participants) | 24 | 24 | 26 | 22 | 18 | 20 | 27 | 30
  252 Days after 1st Vaccine | 2.1 | 2.1 | 2.1 | 2.1 | 2.1 | 2.1 | 2.1 | 1.0
  365 Days after 1st Vaccine: number analyzed (Participants) | 22 | 23 | 26 | 23 | 18 | 20 | 27 | 30
  365 Days after 1st Vaccine | 1.0 | 1.0 | 1.0 | 1.0 | 1.0 | 1.0 | 1.0 | 1.0

18. Secondary Outcome: Absolute Values in Concentrations of Vaccine-induced Antibodies to SARS-CoV-2 Antigens Over Time (S-IgM)
Description: Anti-S protein (Spike protein)
Time Frame: Up to 365 Days from 1st dose of vaccination
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Binding Antibody Unit (BAU)/mL
Arm/Group | Vaccine Only | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 300 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 150 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 48 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 12 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 7 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 SC | REGN10933+REGN10987 + Vaccine 600 mg Day 1 SC
Number analyzed (Participants) | 42 | 26 | 26 | 26 | 28 | 24 | 24 | 32 | 32
Binding Antibody Unit (BAU)/mL
  Baseline: number analyzed (Participants) | 41 | 26 | 26 | 26 | 28 | 24 | 23 | 32 | 32
  Baseline | 5.1 (5.6) | 5.7 (6.6) | 7.1 (9.6) | 5.7 (6.3) | 3.9 (2.9) | 4.8 (3.5) | 4.3 (2.9) | 3.7 (2.0) | 4.3 (3.7)
  6 Days after 1st Vaccine: number analyzed (Participants) | 5 | 0 | 0 | 0 | 0 | 0 | 24 | 0 | 0
  6 Days after 1st Vaccine | 5.0 (2.6) |  |  |  |  |  | 10.0 (21.3) |  |
  14 Days after 1st Vaccine: number analyzed (Participants) | 42 | 26 | 25 | 25 | 28 | 24 | 24 | 31 | 32
  14 Days after 1st Vaccine | 82.1 (84.1) | 50.1 (61.0) | 32.2 (33.4) | 53.8 (99.1) | 579.5 (2919.4) | 21.4 (21.8) | 57.9 (56.6) | 535.1 (2773.1) | 53.8 (133.3)
  28 Days after 1st Vaccine | 52.6 (48.3) | 24.3 (37.2) | 18.7 (28.8) | 23.0 (37.6) | 56.0 (187.7) | 41.4 (136.9) | 34.3 (34.7) | 55.1 (151.0) | 23.4 (52.6)
  42 Days after 1st Vaccine: number analyzed (Participants) | 41 | 25 | 26 | 26 | 28 | 21 | 20 | 32 | 31
  42 Days after 1st Vaccine | 86.3 (90.0) | 57.2 (90.2) | 31.1 (29.5) | 30.4 (26.3) | 604.2 (2914.7) | 66.2 (85.5) | 61.4 (57.3) | 65.5 (111.5) | 42.8 (47.5)
  56 Days after 1st Vaccine: number analyzed (Participants) | 41 | 24 | 26 | 26 | 28 | 22 | 22 | 32 | 31
  56 Days after 1st Vaccine | 50.3 (58.4) | 28.1 (44.0) | 17.8 (20.9) | 14.2 (10.6) | 47.7 (96.6) | 32.3 (39.8) | 42.2 (43.1) | 40.3 (74.5) | 25.9 (29.1)
  168 Days after 1st Vaccine: number analyzed (Participants) | 40 | 24 | 25 | 26 | 25 | 22 | 21 | 31 | 31
  168 Days after 1st Vaccine | 10.4 (9.6) | 7.0 (6.4) | 8.8 (12.4) | 9.7 (14.0) | 16.6 (21.9) | 11.5 (13.4) | 12.1 (8.5) | 7.0 (10.6) | 5.9 (4.8)
  252 Days after 1st Vaccine: number analyzed (Participants) | 37 | 24 | 24 | 26 | 22 | 18 | 20 | 27 | 30
  252 Days after 1st Vaccine | 13.1 (13.9) | 9.6 (6.9) | 10.2 (11.0) | 9.3 (6.8) | 19.9 (45.7) | 11.7 (13.4) | 14.1 (18.5) | 38.4 (147.4) | 15.7 (19.1)
  365 Days after 1st Vaccine: number analyzed (Participants) | 37 | 22 | 23 | 26 | 23 | 18 | 20 | 27 | 30
  365 Days after 1st Vaccine | 8.8 (7.6) | 8.9 (6.4) | 9.5 (9.9) | 8.3 (6.9) | 13.0 (20.4) | 8.0 (6.6) | 13.1 (18.6) | 9.3 (10.0) | 12.5 (13.1)

19. Secondary Outcome: Relative Difference Expressed as a Percent in Concentrations of Vaccine-induced Antibodies to SARS-CoV-2 Antigens Over Time (S-IgM)
Description: Anti-S protein (Spike protein) Relative difference is calculated as: [(LS Geometric Mean Active Arm - LS Geometric Mean Vaccine Alone Arm) / LS Geometric Mean Vaccine Alone Arm] x 100%
Time Frame: Up to 365 Days from 1st dose of vaccination
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 300 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 150 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 48 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 12 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 7 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 SC | REGN10933+REGN10987 + Vaccine 600 mg Day 1 SC
Number analyzed (Participants) | 26 | 26 | 26 | 28 | 24 | 24 | 32 | 32
Percent
  Baseline: number analyzed (Participants) | 26 | 26 | 26 | 28 | 24 | 23 | 32 | 32
  Baseline | 8.9 [-16.7 to 42.4] | 14.7 [-12.4 to 50.1] | 6.3 [-18.7 to 39.1] | -12.1 [-32.4 to 14.3] | 3.9 [-21.1 to 36.9] | -7.3 [-29.9 to 22.6] | -13.3 [-32.7 to 11.6] | -5.8 [-26.9 to 21.5]
  6 Days after 1st Vaccine: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  14 Days after 1st Vaccine: number analyzed (Participants) | 26 | 25 | 25 | 28 | 24 | 24 | 31 | 32
  14 Days after 1st Vaccine | -42.1 [-69.6 to 10.2] | -58.9 [-78.6 to -21.0] | -60.1 [-79.2 to -23.3] | -54.7 [-75.9 to -15.0] | -66.8 [-82.8 to -35.6] | -21.8 [-59.6 to 51.5] | -40.2 [-67.5 to 10.3] | -44.7 [-69.9 to 1.8]
  28 Days after 1st Vaccine | -56.7 [-76.4 to -20.4] | -69.2 [-83.3 to -43.4] | -64.6 [-80.7 to -35.0] | -50.2 [-72.5 to -9.8] | -61.6 [-79.4 to -28.4] | -31.7 [-63.4 to 27.4] | -52.7 [-73.3 to -16.3] | -58.7 [-76.8 to -26.7]
  42 Days after 1st Vaccine: number analyzed (Participants) | 25 | 26 | 26 | 28 | 21 | 20 | 32 | 31
  42 Days after 1st Vaccine | -32.5 [-60.5 to 15.2] | -63.0 [-78.2 to -37.1] | -56.9 [-74.6 to -26.8] | -7.5 [-44.8 to 55.2] | -19.2 [-54.1 to 42.4] | -21.1 [-55.6 to 40.1] | -46.7 [-67.6 to -12.3] | -43.7 [-66.1 to -6.7]
  56 Days after 1st Vaccine: number analyzed (Participants) | 24 | 26 | 26 | 28 | 22 | 22 | 32 | 31
  56 Days after 1st Vaccine | -37.3 [-63.3 to 6.9] | -61.7 [-77.3 to -35.5] | -62.8 [-77.9 to -37.3] | -20.3 [-52.1 to 32.7] | -34.4 [-62.1 to 13.7] | -14.4 [-50.6 to 48.2] | -45.1 [-66.4 to -10.3] | -39.3 [-63.1 to -0.1]
  168 Days after 1st Vaccine: number analyzed (Participants) | 24 | 25 | 26 | 25 | 22 | 21 | 31 | 31
  168 Days after 1st Vaccine | -29.0 [-53.6 to 8.8] | -33.0 [-56.1 to 2.1] | -19.5 [-46.9 to 22.0] | 9.4 [-28.2 to 66.7] | -14.8 [-45.0 to 32.2] | 17.4 [-24.8 to 83.2] | -37.2 [-57.7 to -6.7] | -35.9 [-57.0 to -4.6]
  252 Days after 1st Vaccine: number analyzed (Participants) | 24 | 24 | 26 | 22 | 18 | 20 | 27 | 30
  252 Days after 1st Vaccine | -19.7 [-51.3 to 32.5] | -31.0 [-58.2 to 14.0] | -21.1 [-51.6 to 28.7] | -22.1 [-53.5 to 30.5] | -17.5 [-52.4 to 42.9] | -3.1 [-43.0 to 64.6] | -4.5 [-41.2 to 55.0] | -2.6 [-39.3 to 56.3]
  365 Days after 1st Vaccine: number analyzed (Participants) | 22 | 23 | 26 | 23 | 18 | 20 | 27 | 30
  365 Days after 1st Vaccine | 4.0 [-33.6 to 62.7] | -1.3 [-36.6 to 53.7] | -5.7 [-38.4 to 44.3] | 1.2 [-35.0 to 57.5] | -9.5 [-43.9 to 46.0] | 5.6 [-33.4 to 67.5] | -3.0 [-36.4 to 47.8] | 27.1 [-15.8 to 91.9]

20. Secondary Outcome: Fold Change of Concentrations of Vaccine-induced Antibodies to SARS-CoV-2 Antigens Over Time (S-IgM)
Description: Anti-S protein (Spike protein) Fold Change based on medians = (median value in vaccine only arm / median value in the active arm)
Time Frame: Up to 365 Days from 1st dose of vaccination
Population: as for outcome 3
Measure: Number; unit: Fold Change
Arm/Group | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 300 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 150 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 48 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 12 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 7 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 SC | REGN10933+REGN10987 + Vaccine 600 mg Day 1 SC
Number analyzed (Participants) | 26 | 26 | 26 | 28 | 24 | 24 | 32 | 32
Fold Change
  Baseline: number analyzed (Participants) | 26 | 26 | 26 | 28 | 24 | 23 | 32 | 32
  Baseline | 1.0 | 1.0 | 1.0 | 1.0 | 1.0 | 1.0 | 1.0 | 1.0
  6 Days after 1st Vaccine: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 24 | 0 | 0
  6 Days after 1st Vaccine |  |  |  |  |  | 1.0 |  |
  14 Days after 1st Vaccine: number analyzed (Participants) | 26 | 25 | 25 | 28 | 24 | 24 | 31 | 32
  14 Days after 1st Vaccine | 2.1 | 2.4 | 2.8 | 3.2 | 2.9 | 1.1 | 3.0 | 2.0
  28 Days after 1st Vaccine | 3.6 | 5.2 | 4.5 | 3.3 | 4.9 | 1.9 | 3.7 | 3.7
  42 Days after 1st Vaccine: number analyzed (Participants) | 25 | 26 | 26 | 28 | 21 | 20 | 32 | 31
  42 Days after 1st Vaccine | 2.2 | 2.4 | 2.6 | 1.4 | 1.9 | 1.3 | 2.9 | 2.0
  56 Days after 1st Vaccine: number analyzed (Participants) | 24 | 26 | 26 | 28 | 22 | 22 | 32 | 31
  56 Days after 1st Vaccine | 1.7 | 2.2 | 2.0 | 1.1 | 1.4 | 1.2 | 1.8 | 1.3
  168 Days after 1st Vaccine: number analyzed (Participants) | 24 | 25 | 26 | 25 | 22 | 21 | 31 | 31
  168 Days after 1st Vaccine | 2.7 | 2.7 | 1.8 | 1.3 | 2.7 | 0.9 | 2.7 | 2.7
  252 Days after 1st Vaccine: number analyzed (Participants) | 24 | 24 | 26 | 22 | 18 | 20 | 27 | 30
  252 Days after 1st Vaccine | 1.0 | 3.2 | 1.4 | 3.2 | 1.1 | 1.0 | 1.1 | 1.1
  365 Days after 1st Vaccine: number analyzed (Participants) | 22 | 23 | 26 | 23 | 18 | 20 | 27 | 30
  365 Days after 1st Vaccine | 0.9 | 1.0 | 0.9 | 2.2 | 2.2 | 2.2 | 1.1 | 0.9

21. Secondary Outcome: 50% Inhibitory Dilution (ID50) Titers of Vaccine-induced Neutralizing Antibodies to SARS-CoV-2 S Protein Assessed Over Time After the First Dose of Moderna mRNA-1273 Vaccine
Time Frame: Up to 365 Days from 1st dose of vaccination
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Titer
Arm/Group | Vaccine Only | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 300 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 150 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 48 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 12 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 7 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 SC | REGN10933+REGN10987 + Vaccine 600 mg Day 1 SC
Number analyzed (Participants) | 42 | 26 | 26 | 26 | 28 | 24 | 24 | 32 | 32
Titer
  Baseline | 40.0 (0.0) | 40.0 (0.0) | 40.0 (0.0) | 40.0 (0.0) | 40.0 (0.0) | 40.0 (0.0) | 40.0 (0.0) | 40.0 (0.0) | 40.0 (0.0)
  6 Days: number analyzed (Participants) | 5 | 0 | 0 | 0 | 0 | 0 | 24 | 0 | 0
  6 Days | 40.0 (0.0) |  |  |  |  |  | 827.8 (3859.4) |  |
  14 Days: number analyzed (Participants) | 42 | 26 | 25 | 25 | 28 | 24 | 24 | 31 | 32
  14 Days | 928.4 (4600.0) | 518.7 (1446.0) | 81.0 (59.9) | 84.2 (78.1) | 2686.8 (9365.3) | 780.4 (2955.9) | 1847.5 (6787.1) | 93.3 (78.8) | 1325.2 (6386.1)
  28 Days | 640.5 (2173.9) | 499.8 (1420.1) | 136.2 (169.8) | 177.7 (581.6) | 3887.0 (16628.4) | 631.3 (1955.2) | 785.6 (2134.7) | 113.7 (102.0) | 1108.3 (5103.2)
  42 Days: number analyzed (Participants) | 41 | 25 | 26 | 26 | 28 | 21 | 20 | 32 | 31
  42 Days | 4391.0 (4567.2) | 2623.7 (2216.8) | 1322.6 (1198.8) | 1284.8 (1434.1) | 6926.8 (14487.0) | 3744.3 (4066.7) | 4351.9 (4553.9) | 1418.2 (1414.8) | 2167.2 (5160.7)
  56 Days: number analyzed (Participants) | 41 | 24 | 26 | 26 | 28 | 22 | 22 | 32 | 31
  56 Days | 2594.9 (1981.5) | 1818.6 (2365.8) | 780.8 (771.1) | 716.1 (664.9) | 4922.8 (11157.3) | 2422.2 (2882.7) | 2576.8 (2736.1) | 980.8 (1015.1) | 1549.5 (4334.1)
  168 Days: number analyzed (Participants) | 40 | 24 | 25 | 26 | 25 | 22 | 21 | 31 | 31
  168 Days | 2889.5 (3890.9) | 1756.4 (2759.0) | 649.4 (791.1) | 1670.2 (2774.3) | 3316.2 (4137.5) | 1007.5 (871.8) | 2968.4 (3399.8) | 1261.4 (2139.7) | 974.6 (1124.6)
  252 Days: number analyzed (Participants) | 38 | 24 | 24 | 26 | 22 | 18 | 20 | 28 | 30
  252 Days | 10110.8 (11107.8) | 3815.0 (4058.1) | 2712.6 (2898.7) | 4891.0 (5258.5) | 4844.8 (6960.8) | 6491.6 (12406.5) | 7311.4 (8802.4) | 7034.7 (9548.7) | 5041.1 (6443.0)
  365 Days: number analyzed (Participants) | 37 | 22 | 23 | 26 | 23 | 18 | 20 | 27 | 30
  365 Days | 7250.9 (6902.0) | 7184.3 (6172.6) | 3934.6 (3800.0) | 4408.0 (3941.0) | 7070.1 (9060.8) | 13175.9 (26414.2) | 4949.7 (4445.6) | 6287.3 (6023.3) | 7174.4 (7753.8)

22. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) Throughout the Study
Time Frame: Up to 401 Days
Population: The safety analysis set (SAF) includes all randomized subjects who have been vaccinated with at least one dose or received any study drug; it is based on the treatment received (as treated).
Measure: Number; unit: Participants
Arm/Group | Vaccine Only | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 300 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 150 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 48 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 12 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 7 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 SC | REGN10933+REGN10987 + Vaccine 600 mg Day 1 SC
Number analyzed (Participants) | 48 | 28 | 29 | 28 | 33 | 31 | 26 | 35 | 35
Participants | 22 | 13 | 16 | 17 | 15 | 16 | 13 | 16 | 23

23. Secondary Outcome: Number of Participants With Treatment-emergent Serious Adverse Events (SAEs) Throughout the Study
Time Frame: Up to 401 Days
Population: as for outcome 22
Measure: Number; unit: Participants
Arm/Group | Vaccine Only | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 300 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 150 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 48 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 12 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 7 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 SC | REGN10933+REGN10987 + Vaccine 600 mg Day 1 SC
Number analyzed (Participants) | 48 | 28 | 29 | 28 | 33 | 31 | 26 | 35 | 35
Participants | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0

24. Secondary Outcome: Number of Participants With Infusion-related Reactions (Grade ≥2) to REGN10933+REGN10987
Time Frame: Through Day 4 post-infusion
Population: as for outcome 22
Measure: Number; unit: Participants
Arm/Group | Vaccine Only | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 300 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 150 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 48 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 12 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 7 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 SC | REGN10933+REGN10987 + Vaccine 600 mg Day 1 SC
Number analyzed (Participants) | 48 | 28 | 29 | 28 | 33 | 31 | 26 | 35 | 35
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

25. Secondary Outcome: Number of Participants With Injection Site Reactions (Grade ≥3) to REGN10933+REGN10987
Time Frame: Through Day 4 post-infusion
Population: as for outcome 22
Measure: Number; unit: Participants
Arm/Group | Vaccine Only | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 300 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 150 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 48 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 12 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 7 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 SC | REGN10933+REGN10987 + Vaccine 600 mg Day 1 SC
Number analyzed (Participants) | 48 | 28 | 29 | 28 | 33 | 31 | 26 | 35 | 35
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

26. Secondary Outcome: Number of Participants With Injection Site Reactions (Grade ≥3) to Moderna mRNA-1273 Vaccine
Time Frame: Through Day 4 post-infusion
Population: as for outcome 22
Measure: Number; unit: Participants
Arm/Group | Vaccine Only | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 300 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 150 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 48 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 12 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 7 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 SC | REGN10933+REGN10987 + Vaccine 600 mg Day 1 SC
Number analyzed (Participants) | 48 | 28 | 29 | 28 | 33 | 31 | 26 | 35 | 35
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

27. Secondary Outcome: Number of Participants With Hypersensitivity Reactions (Grade ≥2) to REGN10933+REGN10987 or Each Dose of Moderna mRNA-1273 Vaccine
Description: Grade 2 - characterized by an adverse local or general response from exposure and oral intervention indicated Grade 3 - hospitalization indicated and intravenous response required Grade 4 - Life Threatening consequence and urgent intervention indicated Grade 5 - Death
Time Frame: Through Day 29 post-infusion or post-injection
Population: The safety analysis set (SAF) includes all randomized subjects who have been vaccinated with at least one dose or received any study drug; it is based on the treatment received (as treated). Groups assessment based on time and route of administration
Measure: Number; unit: Participants
Arm/Group | Vaccine Only | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 300 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 150 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 48 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 12 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 7 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 SC | REGN10933+REGN10987 + Vaccine 600 mg Day 1 SC
Number analyzed (Participants) | 48 | 28 | 29 | 28 | 33 | 31 | 26 | 35 | 35
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

28. Secondary Outcome: Concentrations of REGN10933 in Serum Over Time
Time Frame: Up to 182 Days
Population: The pharmacokinetics (PK) analysis sets (PKAS) are defined for each study drug separately and includes all subjects who received any study drug and who had at least 1 non-missing result following the first dose of the respective study drug.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 300 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 150 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 48 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 12 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 7 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 SC | REGN10933+REGN10987 + Vaccine 600 mg Day 1 SC
Number analyzed (Participants) | 28 | 29 | 28 | 33 | 31 | 26 | 35 | 35
mg/L
  0 Days (Pre-dose): number analyzed (Participants) | 27 | 28 | 28 | 33 | 17 | 26 | 35 | 35
  0 Days (Pre-dose) | 0.0219 (0.114) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5.12 (26.1) | 0 (0) | 0 (0)
  0 Days (End of Infusion): number analyzed (Participants) | 27 | 28 | 28 | 31 | 16 | 26 | 35 | 35
  0 Days (End of Infusion) | 145 (40.8) | 40.5 (16.2) | 26.8 (16.9) | 7.84 (4.28) | 1.84 (0.593) | 140 (54.4) | 0.527 (0.966) | 0.0765 (0.160)
  8 Days: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 26 | 0 | 0
  8 Days |  |  |  |  |  | 63.7 (11.7) |  |
  14 Days: number analyzed (Participants) | 26 | 26 | 27 | 32 | 17 | 0 | 34 | 35
  14 Days | 46.8 (11.3) | 12.7 (3.79) | 8.30 (3.94) | 2.62 (1.44) | 0.536 (0.229) |  | 39.4 (11.5) | 20.4 (7.48)
  22 Days: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 26 | 0 | 0
  22 Days |  |  |  |  |  | 39.1 (10.9) |  |
  28 Days: number analyzed (Participants) | 26 | 26 | 26 | 30 | 17 | 0 | 34 | 35
  28 Days | 29.5 (9.89) | 8.24 (3.02) | 5.12 (2.28) | 1.76 (1.13) | 0.354 (0.150) |  | 26.0 (8.04) | 14.7 (6.25)
  36 Days: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 22 | 0 | 0
  36 Days |  |  |  |  |  | 27.7 (7.80) |  |
  42 Days: number analyzed (Participants) | 26 | 26 | 27 | 31 | 17 | 0 | 34 | 34
  42 Days | 18.7 (7.98) | 5.38 (2.40) | 3.35 (1.71) | 1.19 (0.861) | 0.237 (0.114) |  | 17.5 (6.30) | 9.77 (5.01)
  50 Days: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 24 | 0 | 0
  50 Days |  |  |  |  |  | 19.3 (5.45) |  |
  56 Days: number analyzed (Participants) | 25 | 29 | 27 | 31 | 13 | 0 | 34 | 34
  56 Days | 13.4 (5.87) | 3.51 (1.78) | 2.10 (1.14) | 0.754 (0.569) | 0.131 (0.142) |  | 11.6 (5.04) | 6.70 (3.77)
  70 Days: number analyzed (Participants) | 24 | 26 | 27 | 31 | 15 | 0 | 0 | 0
  70 Days | 9.98 (6.06) | 2.34 (1.33) | 1.42 (0.804) | 0.522 (0.456) | 0.0105 (0.0408) |  |  |
  162 Days: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 23 | 0 | 0
  162 Days |  |  |  |  |  | 1.38 (1.00) |  |
  168 Days: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 33 | 34
  168 Days |  |  |  |  |  |  | 0.891 (0.712) | 0.615 (0.797)
  182 Days: number analyzed (Participants) | 24 | 25 | 27 | 27 | 16 | 0 | 0 | 0
  182 Days | 0.898 (1.06) | 0.180 (0.212) | 0.137 (0.356) | 0.00693 (0.0360) | 0 (0) |  |  |

29. Secondary Outcome: Concentrations of REGN10987 in Serum Over Time
Time Frame: Up to 182 Days
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 300 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 150 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 48 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 12 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 7 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 SC | REGN10933+REGN10987 + Vaccine 600 mg Day 1 SC
Number analyzed (Participants) | 28 | 29 | 28 | 33 | 31 | 26 | 35 | 35
mg/L
  0 Days (Pre-dose): number analyzed (Participants) | 27 | 28 | 28 | 33 | 17 | 26 | 35 | 35
  0 Days (Pre-dose) | 0.0223 (0.116) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6.00 (30.6) | 0 (0) | 0.00577 (0.0341)
  0 Days (End of Infusion): number analyzed (Participants) | 27 | 28 | 28 | 31 | 16 | 26 | 35 | 35
  0 Days (End of Infusion) | 144 (42.5) | 39.6 (15.5) | 28.9 (26.7) | 8.60 (5.10) | 1.91 (0.687) | 150 (58.0) | 0.580 (0.777) | 0.232 (0.614)
  8 Days: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 26 | 0 | 0
  8 Days |  |  |  |  |  | 61.6 (12.0) |  |
  14 Days: number analyzed (Participants) | 26 | 26 | 27 | 32 | 17 | 0 | 34 | 35
  14 Days | 40.0 (11.2) | 11.2 (3.41) | 7.20 (3.09) | 2.33 (1.37) | 0.438 (0.226) |  | 33.8 (9.51) | 18.0 (6.15)
  22 Days: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 26 | 0 | 0
  22 Days |  |  |  |  |  | 35.0 (10.5) |  |
  28 Days: number analyzed (Participants) | 26 | 25 | 26 | 30 | 17 | 0 | 34 | 35
  28 Days | 23.8 (9.92) | 6.87 (2.84) | 4.19 (1.95) | 1.46 (0.968) | 0.263 (0.189) |  | 21.0 (6.95) | 12.1 (5.92)
  36 Days: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 22 | 0 | 0
  36 Days |  |  |  |  |  | 22.2 (6.56) |  |
  42 Days: number analyzed (Participants) | 26 | 26 | 27 | 31 | 17 | 0 | 34 | 34
  42 Days | 13.7 (6.86) | 4.00 (2.02) | 2.54 (1.35) | 0.868 (0.641) | 0.138 (0.147) |  | 13.3 (6.11) | 7.71 (4.42)
  50 Days: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 24 | 0 | 0
  50 Days |  |  |  |  |  | 14.5 (4.09) |  |
  56 Days: number analyzed (Participants) | 25 | 26 | 27 | 31 | 13 | 0 | 34 | 34
  56 Days | 9.23 (4.97) | 2.51 (1.48) | 1.55 (0.903) | 0.507 (0.453) | 0.0776 (0.138) |  | 8.02 (3.99) | 4.86 (3.07)
  70 Days: number analyzed (Participants) | 24 | 29 | 27 | 31 | 15 | 0 | 0 | 0
  70 Days | 6.51 (4.53) | 1.57 (1.04) | 0.993 (0.630) | 0.306 (0.344) | 0.0115 (0.0444) |  |  |
  162 Days: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 23 | 0 | 0
  162 Days |  |  |  |  |  | 0.566 (0.560) |  |
  168 Days: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 33 | 34
  168 Days |  |  |  |  |  |  | 0.347 (0.378) | 0.251 (0.465)
  182 Days: number analyzed (Participants) | 24 | 25 | 27 | 27 | 16 | 0 | 0 | 0
  182 Days | 0.400 (0.617) | 0.0401 (0.124) | 0.0408 (0.179) | 0 (0) | 0 (0) |  |  |

30. Secondary Outcome: Immunogenicity, as Measured by Anti-drug Antibodies (ADA) to REGN10987
Time Frame: Up to Day 183
Population: as for outcome 28
Measure: Number; unit: Percent of Participants
Arm/Group | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 300 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 150 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 48 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 12 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 7 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 SC | REGN10933+REGN10987 + Vaccine 600 mg Day 1 SC
Number analyzed (Participants) | 27 | 27 | 27 | 30 | 30 | 23 | 34 | 35
Percent of Participants
  Negative | 48.1 | 55.6 | 44.4 | 46.7 | 56.7 | 56.5 | 55.9 | 57.1
  Pre-Existing Immunoreactivity | 7.4 | 0 | 3.7 | 3.3 | 3.3 | 8.7 | 0 | 5.7
  Treatment-Boosted Response | 0 | 0 | 0 | 3.3 | 0 | 0 | 2.9 | 0

31. Secondary Outcome: Immunogenicity, as Measured by Anti-drug Antibodies (ADA) to REGN10933
Time Frame: Up to Day 183
Population: The AAS are defined for each study drug separately and include all treated participants who received any amount of study drug (active [SAF]) and had at least 1 non-missing ADA result of respective analyte following the first dose of study drug.
Measure: Number; unit: Percent of Participants
Arm/Group | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 300 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 150 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 48 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 12 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 7 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 SC | REGN10933+REGN10987 + Vaccine 600 mg Day 1 SC
Number analyzed (Participants) | 27 | 27 | 27 | 30 | 30 | 23 | 34 | 35
Percent of Participants
  Negative | 66.7 | 59.3 | 44.4 | 30.0 | 36.7 | 91.3 | 70.6 | 62.9
  Pre-Existing Immunoreactivity | 0 | 3.7 | 3.7 | 6.7 | 0 | 0 | 0 | 0
  Treatment-Boosted Response | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

32. Secondary Outcome: Immunogenicity, as Measured by Neutralizing Antibodies (NAb) to REGN10987
Time Frame: Up to Day 183
Population: The NAbS are defined for each study drug separately and comprises all treated participants (active) that were included in the AAS and tested negative at all ADA sampling times or tested positive at 1 or more postdose ADA sampling times and had at least 1 non-missing postdose NAb result (imputed or analysis result).
Measure: Count of Participants; unit: Participants
Arm/Group | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 300 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 150 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 48 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 12 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 7 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 SC | REGN10933+REGN10987 + Vaccine 600 mg Day 1 SC
Number analyzed (Participants) | 27 | 27 | 27 | 30 | 30 | 23 | 34 | 35
Participants
  NAb Negative | 16 | 12 | 16 | 17 | 20 | 15 | 24 | 22
  NAb Positive | 11 | 6 | 11 | 13 | 10 | 8 | 10 | 13

33. Secondary Outcome: Immunogenicity, as Measured by Neutralizing Antibodies (NAb) to REGN10933
Time Frame: Up to Day 183
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 300 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 150 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 48 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 12 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 7 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 SC | REGN10933+REGN10987 + Vaccine 600 mg Day 1 SC
Number analyzed (Participants) | 27 | 27 | 27 | 30 | 30 | 23 | 34 | 35
Participants
  NAb Negative | 27 | 25 | 26 | 22 | 23 | 21 | 32 | 32
  Nab Positive | 0 | 2 | 1 | 8 | 7 | 2 | 2 | 3

ADVERSE EVENTS:
Time Frame: Up to 401 Days
Groups:
- Vaccine Only Total All: Vaccine only, no study intervention
Arm/Group | Vaccine Only Total All | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 300 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 150 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 SC | REGN10933+REGN10987 + Vaccine 600 mg Day 1 SC | REGN10933+REGN10987 + Vaccine 48 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 12 mg Day 1 IV | REGN10933+REGN10987 + Vaccine 1200 mg Day 7 IV
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/28 | 0/29 | 0/28 | 0/35 | 0/35 | 0/33 | 0/31 | 1/26
Serious Adverse Events (participants affected / at risk) | 2/48 | 0/28 | 0/29 | 0/28 | 1/35 | 0/35 | 0/33 | 0/31 | 2/26
Other Adverse Events (participants affected / at risk) | 11/48 | 13/28 | 9/29 | 14/28 | 15/35 | 23/35 | 12/33 | 14/31 | 9/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vaccine Only Total All (N=48) | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 IV (N=28) | REGN10933+REGN10987 + Vaccine 300 mg Day 1 IV (N=29) | REGN10933+REGN10987 + Vaccine 150 mg Day 1 IV (N=28) | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 SC (N=35) | REGN10933+REGN10987 + Vaccine 600 mg Day 1 SC (N=35) | REGN10933+REGN10987 + Vaccine 48 mg Day 1 IV (N=33) | REGN10933+REGN10987 + Vaccine 12 mg Day 1 IV (N=31) | REGN10933+REGN10987 + Vaccine 1200 mg Day 7 IV (N=26)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic foot infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vaccine Only Total All (N=48) | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 IV (N=28) | REGN10933+REGN10987 + Vaccine 300 mg Day 1 IV (N=29) | REGN10933+REGN10987 + Vaccine 150 mg Day 1 IV (N=28) | REGN10933+REGN10987 + Vaccine 1200 mg Day 1 SC (N=35) | REGN10933+REGN10987 + Vaccine 600 mg Day 1 SC (N=35) | REGN10933+REGN10987 + Vaccine 48 mg Day 1 IV (N=33) | REGN10933+REGN10987 + Vaccine 12 mg Day 1 IV (N=31) | REGN10933+REGN10987 + Vaccine 1200 mg Day 7 IV (N=26)
COVID-19 (Infections and infestations) | 5 (5) | 7 (8) | 3 (3) | 3 (4) | 7 (7) | 6 (6) | 0 (0) | 6 (6) | 3 (3)
Asymptomatic COVID-19 (Infections and infestations) | 3 (3) | 2 (2) | 4 (4) | 9 (9) | 6 (6) | 7 (7) | 4 (4) | 4 (4) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (4) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 4 (5) | 3 (3) | 3 (3) | 1 (2)
Injection site reaction (General disorders) | 2 (2) | 2 (3) | 1 (1) | 1 (2) | 7 (8) | 12 (17) | 1 (1) | 1 (1) | 5 (6)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 2 (2) | 1 (1) | 2 (3)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2022-01-28): https://cdn.clinicaltrials.gov/large-docs/78/NCT04852978/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-23): https://cdn.clinicaltrials.gov/large-docs/78/NCT04852978/SAP_001.pdf